#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for a 24- week randomised, double-blind and placebo-controlled study to evaluate the efficacy and safety of 62.5 mcg Umeclidinium Inhalation Powder delivered once-daily via a Novel Dry Powder Inhaler in subjects with Chronic Obstructive Pulmonary Disease |
|---|---|---|
| <b>Compound Number</b> | : | GSK573719 |
| <b>Effective Date</b> | : | 26-DEC-2017 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be performed on all subjects enrolled from China and Korea and on the subjects enrolled in China alone: A China subgroup analysis for Protocol AC4117410.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### RAP Author(s):

| Author | Date |
|----------------------------------------------------------|-------------|
| Senior Statistician, Statistics & Programming, R&D China | 26-DEC-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

#### The GlaxoSmithKline group of companies

#### **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Principal Statistician, Clinical Statistics | 23-DEC-2017 | E-mail approved |
| Clinical Research Physician, R&D China | 26-DEC-2017 | E-mail approved |
| Senior Clinical Research Physician, R&D China | 04-DEC-2017 | E-mail approved |
| Senior Programmer, R&D China | 26-DEC-2017 | E-mail approved |
| Senior Study Manager, R&D China | 25-DEC-2017 | E-mail approved |
| Senior Clinical Data Scientist, R&D China | 26-DEC-2017 | E-mail approved |

#### **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Associate Director, Statistics & Programming, R&D China | 25-DEC-2017 | E-mail approved |

#### **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPC | RTING & | ANALYSIS PLAN SYNPOSIS | 6 |
| 2. | CLIMAN | ANDV OF | KEY PROTOCOL INFORMATION | Ω |
| ۷. | 2.1. | _ | s to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | | bjective(s) and Endpoint(s) | |
| | 2.3. | | esign | |
| | 2.4. | | al Hypotheses | |
| | | | · · | |
| 3. | PLAN | | LYSES | |
| | 3.1. | | Analyses | |
| | 3.2. | Final An | alyses | 11 |
| 4. | ANAL | YSIS POF | PULATIONS | 11 |
| | 4.1. | Protocol | Deviations | 13 |
| 5. | CONS | NDEDATI | ONS FOR DATA ANALYSES AND DATA HANDLING | |
| Ο. | | | ONS FOR DATA ANALTSES AND DATA HANDLING<br>S | 14 |
| ^ | OTUD | V DODLII | ATION ANALYOFO | 4.5 |
| 6. | | | ATION ANALYSES | |
| | 6.1. | Overvie | w of Planned Analyses | 15 |
| 7. | | | TISTICAL ANALYSES | |
| | 7.1. | | Efficacy Analyses | |
| | | 7.1.1. | Overview of Planned Primary Efficacy Analyses | |
| | | 7.1.2. | Planned Primary Efficacy Statistical Analyses | 18 |
| | | 7.1.3. | Planned Missing Data Sensitivity Statistical Analyses for Trough FEV1 | 20 |
| | 7.2. | Seconda | ary Efficacy Analyses | |
| | 1.2. | 7.2.1. | Overview of Planned Secondary Efficacy Analyses | |
| | | 7.2.2. | Planned Secondary Efficacy Statistical Analyses | |
| | | | 7.2.2.1. 0-6 h Weighted Mean FEV1 on Day 1 | |
| | | | 7.2.2.2. TDI | |
| | 7.3. | Other Ef | fficacy Analyses | |
| | | 7.3.1. | Overview of Planned Other Efficacy Analyses | |
| | | 7.3.2. | Planned Other Efficacy Statistical Analyses | |
| | | | 7.3.2.1. Time to Onset and Time to First COPD | |
| | | | Exacerbation | 24 |
| | | | 7.3.2.2. Proportion Endpoints | |
| | | | 7.3.2.3. Serial FEV1/FVC and Trough FVC | |
| | | | 7.3.2.4. Rescue Salbutamol Use (mean puffs/days) | |
| | 7.4. | Health C | Outcomes Analyses | |
| | | 7.4.1. | Overview of Planned Health Outcomes Analyses | |
| | | 7.4.2. | Planned Health Outcomes Statistical Analyses | |
| 8. | SAFE | TY ΔΝΙΛΙ Υ | YSES | 20 |
| ٥. | 8.1. | | Events Analyses | |
| | 0.1. | 8.1.1. | Overview of Planned Adverse Events Analyses | |
| | 8.2. | _ | Laboratory Analyses | |
| | 0.2. | 8.2.1. | Overview of Planned Clinical Laboratory Analyses | 30 |


| | 8.3. | Other Sa | | <del>?</del> S | |
|---|---|---|---|---|---|
| | | 8.3.1. | Overview o | f Planned Other Safety Analyses | 31 |
| | | 8.3.2. | Planned Sa | afety Statistical Analyses | 32 |
| | | | | , | |
| 9. | REFE | RENCES. | | | 33 |
| 10. | APPE | NDICES | | | 34 |
| | 10.1. | | | Deviation Management and Definitions for Per | |
| | | | | | 35 |
| | | 10.1.1. | | of Data from Modified Intent-to-treat Analyses | |
| | | 10.1.2. | | of Data from Per Protocol Analyses | |
| | | | | clusion/randomisation Criteria Deviations | |
| | | 10.1.2.1 | | ed Checks to Identify Non-medication | 00 |
| | | 10.1.5. | Dovistions | | 26 |
| | | 10 1 1 | | | |
| | 40.0 | 10.1.4. | | ed Checks to Identify Medication Deviations | |
| | 10.2. | | | Events | |
| | 40.0 | 10.2.1. | | efined Time & Events | |
| | 10.3. | | | nent Windows | |
| | 10.4. | | | nt States and Phases | |
| | | 10.4.1. | | Phases | |
| | | 10.4.2. | | States | 43 |
| | | | | Treatment States for Concomitant Medications | |
| | | | | Data | |
| | | | | Treatment States for AE Data | |
| | | | 10.4.2.3. | Treatment States for COPD exacerbation | 44 |
| | 10.5. | Appendix | 5: Data Dis | splay Standards & Handling Conventions | 45 |
| | | 10.5.1. | | tment & Sub-group Display Descriptors | |
| | | 10.5.2. | | efinition & Derivations | |
| | | | 10.5.2.1. | Baseline Definitions | 45 |
| | | | | Derivations and Handling of Missing Baseline | |
| | | | | Data | 45 |
| | | 10.5.3. | | Process & Standards | |
| | 10.6. | | | and Transformed Data | |
| | 10.0. | 10.6.1. | | | |
| | | 10.6.1. | | llation | |
| | | 10.6.2. | , , | ilation | |
| | | 10.6.4. | | ated Quality of Life | |
| | | 10.6.4. | | | |
| | 40.7 | | | wa With day, als O Handling of Missing Date | |
| | 10.7. | | | re Withdrawals & Handling of Missing Data | |
| | | 10.7.1. | | Withdrawals | |
| | | 10.7.2. | | Missing Data | |
| | | | | Handling of Missing Responder | |
| | | | | Handing of Missing Dates | |
| | | | | Handling of Partial Dates | 59 |
| | | | | Handling of Missing Data for Statistical | |
| | | | | Analysis | |
| | 10.8. | Appendix | | of Potential Clinical Importance | |
| | | 10.8.1. | Laboratory | Values | 61 |
| | | 10.8.2. | ECG | | 61 |
| | | 10.8.3. | | | |
| | 10.9. | | • | ter Studies | |
| | 10.10. | | | nation of Covariates, Subgroups & Other Strata | |


#### AC4117410

| 10.11. | Appendix | 11: Multiple Comparisons & Multiplicity | 64 |
|--------|----------|----------------------------------------------------|----|
| 10.12. | Appendix | 12: Model Checking and Diagnostics for Statistical | |
| | Analyses | | 65 |
| | | Statistical Analysis Assumptions | |
| 10.13. | | c 13 – Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 10.14. | | c 14: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverable [Priority] | |
| | | Study Population Tables | |
| | | Study Population Figures | |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables | |
| | 10.14.9. | Safety Figures | 90 |
| | | .ICH Listings | |
| | | Non-ICH Listings | |
| 10.15. | | 15: Example Mock Shells for Data Displays | |

#### 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP describes the analysis to be performed on all subjects enrolled from China, Korea and also the subjects enrolled in China alone: a China subgroup analysis for study AC4117410. |
| Protocol | <ul> <li>This RAP is based on the protocol amendment 03 [(Dated: 11/Nov/2015) of<br/>study AC4117410 (GSK Document Number. 2013N159587_03] and eCRF<br/>Version (1.3).</li> </ul> |
| Primary<br>Objective | <ul> <li>Evaluate the efficacy of Umeclidinium Inhalation Powder at 62.5 mcg compared<br/>with placebo when administered once-daily via ELLIPTA™ over a 24-week<br/>treatment period in subjects with COPD</li> </ul> |
| Primary<br>Endpoint | Change from baseline of clinic visit trough (pre-bronchodilator) FEV1 on Treatment Day 169 |
| | Trough FEV1 on Treatment Day 169 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on Treatment Day 168 (i.e. at Week 24). |
| | [Note: This has been altered from the Protocol GSK Document Number 2013N159587_03 where the endpoint was not clarified change from baseline] |
| Study<br>Design | 24-week, phase III multicenter, randomized, double-blind, placebo-controlled, parallel-group study. |
| | Planned total number of approximately 288 randomized subjects will be randomised to UMEC 62.5 mcg and placebo treatment group in a 2:1 ratio. |
| | A total of 10 study clinic visits are planned to be conducted on an outpatient basis but may be less if subjects withdraw from study. |
| | The total duration of subject participation, including follow-up will be approximately 27 weeks. |
| | All subjects will be provided with albuterol/salbutamol for use on an "as-needed" basis throughout the Pre-screen, Run-in and study Treatment periods. |
| Planned<br>Analyses | All decisions regarding final analysis, as defined in this RAP document, will be made prior to Database Freeze (unblinding) of the study data. |
| Analysis<br>Populations | The All Subjects Enrolled Population will be used for reporting subject disposition, AE listing and treatment misallocations listing. |
| | The Screen and Run in Failure population will be used for the tabulation of reasons for screen and run-in failure and for inclusion, exclusion and randomisation criteria failed. |
| | The Modified Intent-to-treat (ITT) Population will constitute the primary population for all data analyses and displays. |
| | The Per Protocol (PP) Population will be used for confirmatory analyses of the primary endpoint only, irrespective of how many subjects are in the PP population. |

| Overview | Key Elements of the RAP |
|---|---|
| Hypothesis | For each test on each efficacy endpoint: |
| | The null hypothesis is that there is no difference between Umeclidinium 62.5 mcg and placebo. |
| | <ul> <li>H₀: T₁ - T₂ = 0</li> <li>The alternative hypothesis is there is a difference between Umeclidinium 62.5 mcg and placebo.</li> </ul> |
| | $H_1: T_1 - T_2 \neq 0$ |
| Primary<br>Analyses | The primary endpoint of change from baseline trough in FEV1 on Day 169 will be analysed for the Modified Intent-to-treat Population using a mixed model repeated measures (MMRM) analysis, including trough FEV1 recorded at each of Days 2, 28, 56, 84, 112, 168 and 169. |
| Secondary<br>Analyses | The analysis of the mean Transition Dyspnea Index (TDI) focal score on Days 28, 84 and 168 will use the same methodology as that for the primary endpoint. |
| | Weighted mean clinic visit FEV1 over 0 to 6 hours post-dose at Visit 2 (Day 1) will be analysed using analysis of covariance (ANCOVA). |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

#### 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There was one change to the originally planned statistical analysis specified in the protocol amendment 03 (Dated: 11-NOV-2015) of study AC4117410 (GSK Document Number 2013N159587\_03). This change was made so that primary endpoint description is consistent across all documents.

In the following section of the protocol, the primary endpoint is Clinic visit trough (pre-bronchodilator) FEV1 on Treatment Day 169.

PROTOCOL SUMMARY
OBJECTIVE(S) and Endpoints (Section 2)
Efficacy (Section 6.2)
Hypotheses (Section 8.1)
Sample Size Assumptions (Section 8.2.1)

In Efficacy Analyses Section (8.3.5.1), it is clarified that the primary endpoint is change from baseline trough in FEV1 on Day 169.

Actually, the primary endpoint of this study is change from baseline in trough FEV1 on Day 169. The sample size calculation was based on this endpoint. To avoid any confusion, the primary endpoint has been defined as change from baseline in trough FEV1 on Day 169 in this RAP.

#### 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | |
| <ul> <li>To evaluate the</li> </ul> | Primary Efficacy Endpoints: |
| efficacy of<br>Umeclidinium 62.5 | <ul> <li>Change from Baseline of Clinic visit trough (pre-bronchodilator) FEV₁ on<br/>Treatment Day 169</li> </ul> |
| mcg compared<br>with placebo when<br>administrated | Trough FEV <sub>1</sub> on Treatment Day 169 is defined as the mean of the FEV <sub>1</sub> values obtained 23 and 24 hours after dosing on Treatment Day 168 (i.e. at Week 24). |
| once-daily via the | Secondary Efficacy Endpoints: |
| ELLIPTATM over | TDI focal score at Week 24 (Day 168) |
| a 24-week<br>treatment period in | <ul> <li>Weighted mean clinic visit FEV<sub>1</sub> over 0 to 6 hours post-dose at visit 2<br/>(Randomization visit, Day 1)</li> </ul> |
| subjects with<br>COPD | Other Efficacy Endpoints: |
| COPD | Trough FEV <sub>1</sub> and TDI focal score at other time points |
| | Rescue albuterol/salbutamol use (percentage of rescue-free days and puffs/day) |
| | <ul> <li>Time to onset (defined as an increase of 100mL above baseline in FEV<sub>1</sub>)<br/>during 0-6hr post-dose on Treatment Day 1 (Visit 2)</li> </ul> |
| | <ul> <li>Proportion of subjects achieving an increase in FEV₁ of ≥12% and ≥200mL<br/>above baseline at any time during 0 to 6hr post-dose on Treatment Day 1<br/>(Visit 2)</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | <ul> <li>Proportion of subjects achieving an increase in FEV₁ of ≥100mL above<br/>baseline in trough FEV₁</li> </ul> |
| | Serial FEV <sub>1</sub> over 0 to 6 hours post-dose (on Day 1) |
| | Serial and trough Forced Vital Capacity (FVC) |
| | Proportion of responders to TDI. (a responder to TDI will be defined as a subject with TDI score of 1 unit or more) |
| | Time to first COPD exacerbation |
| Secondary Objective | s |
| <ul> <li>To evaluate the</li> </ul> | Incidence of adverse events |
| safety of | Vital signs (pulse rate, systolic and diastolic blood pressure) |
| Umeclidinium 62.5 | 12-lead ECG parameters |
| mcg compared with placebo when administrated once-daily via ELLIPTA over a 24-week treatment period in subjects with COPD | Clinical chemistry and haematology parameters and routine urinalysis |
| <ul> <li>To evaluate</li> </ul> | St. George's Respiratory Questionnaire (SGRQ) |
| health-related | COPD Assessment Test (CAT) |
| quality of life Umeclidinium 62.5 mcg compared with placebo when administrated once-daily via ELLIPTA over a 24-week treatment period in subjects with COPD | Healthcare resource utilisation |

#### 2.3. Study Design



#### 2.4. Statistical Hypotheses

The objective of this study is to assess the efficacy and safety of 24 weeks' treatment with Umeclidinium 62.5 mcg Inhalation Powder compared with placebo, when administered once-daily in subjects with COPD. The primary endpoint is change from baseline of trough FEV1 at Day 169. The comparisons of interest for the primary analysis are Umeclidinium 62.5 mcg vs. placebo.

For each test on each efficacy endpoint, the null hypothesis is that there is no difference between treatment groups.

H0: T1 - T2 = 
$$0$$

The alternative hypothesis is there is a difference between treatment groups.

H1: T1 - T2 
$$\neq$$
 0

#### 3. PLANNED ANALYSES

#### 3.1. Interim Analyses

No interim analysis is planned.

#### 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

Population for analysis to be performed on all subjects enrolled from China and Korea.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Enrolled | Comprise of all subjects, for whom a record exists on the study database, including pre-screen/screen failures and any subject who was not screened but experienced an SAE between the date of informed consent and the planned date of the Screening Visit. | Reporting subject disposition, AE listing and treatment misallocations listing |
| Screen and<br>Run in Failure | Comprise of all subjects in the All<br>Subjects Enrolled Population who are<br>recorded as screen failures or run-in<br>failures in the electronic case report<br>form (eCRF) | Tabulation of reasons for<br>screen and run-in failure and<br>for inclusion, exclusion and<br>randomisation criteria failed |
| Modified Intent-<br>To-Treat | Comprise of all subjects randomized to<br>treatment who received at least one<br>dose of randomized study medication in<br>the treatment period. | Constitute the primary population for all data analyses and displays. |
| | Randomized subjects will be assumed to have received study medication unless definitive evidence to the contrary exists. | |
| | Outcomes will be reported according to<br>the randomized treatment allocation. | |
| | All scheduled data collected until the | |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | time of study discontinuation will be included in the Modified Intent-to-treat analysis for subjects who withdraw from the study. | |
| Per-Protocol | Comprise all subjects in the Modified<br>ITT Population who are not identified as<br>full protocol violators. | Confirmatory analyses of the primary efficacy endpoint only, irrespective of how |
| | Subjects identified as partial protocol violators will be included in the PP Population but will have their data excluded from PP analyses from the time of violation onwards. | many subjects are in the PP population. |
| • | The definition of full and partial violations will be included in Section 4.1 (Protocol Deviations) and Appendix 1 (Protocol Deviation Management and Definition for Per-Protocol Population). | |
| | The decision to exclude a subject from<br>the PP Population or a subject's data<br>from PP analyses will be made prior to<br>breaking the blind. | |

Please refer to Appendix 14: List of Data Displays which details the population to be used for each display being generated.

Population for analysis to be performed on subjects enrolled in China alone: a China subgroup analysis.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| China All<br>Subjects Enrolled | Comprise of all subjects as defined in<br>the above table in All Subjects<br>Enrolled population, but will include<br>only those subjects at sites in China. | The same as above table for<br>All Subjects Enrolled<br>Population. |
| China Screen and<br>Run in Failure | Comprise of all subjects as defined in<br>the above table in Screen and Run in<br>Failure population, but will include<br>only those subjects at sites in China | The same as above table for<br>Screen and Run in Failure<br>Population. |
| China Modified<br>Intent-To-Treat | Comprise of all subjects as defined in<br>the above table in Modified Intent-To-<br>Treat Population, but will include only<br>those subjects at sites in China. | The same as above table for Modified Intent-To-Treat Population. |
| China Per-<br>Protocol | Comprise all subjects as defined in<br>the above table in Per-Protocol<br>Population, but will include only those | The same as above table for<br>Per-Protocol Population. |

| Population | Definition / Criteria | Analyses Evaluated |
|------------|-----------------------------|--------------------|
| | subjects at sites in China. | |

Please refer to Appendix 14: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Assessment Windows |
| Section 10.4 | Appendix 4: Treatment States & Phases |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 10.9 | Appendix 9: Multicentre Studies |
| Section 10.10 | Appendix 10: Examination of Covariates and Subgroups |
| Section 10.11 | Appendix 11: Multiple Comparisons and Multiplicity |
| Section 10.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | |
| Section 10.13 | Appendix 13: Abbreviations & Trade Marks |
| Section 10.14 | Appendix 14: List of Data Displays |
| Section 10.15 | Appendix 15: Example Mock Shells for Data Displays |

#### 6. STUDY POPULATION ANALYSES

#### 6.1. Overview of Planned Analyses

The study population analyses will be based on the Modified Intent-To-Treat population for the analysis on all countries overall and on China Modified Intent-To-Treat population for the analysis of China subgroup alone, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays. All the planned study population analyses will be done on all countries overall, and China subgroup alone (with the exception of those displays specified by country).

Table 2 Overview of Planned Study Population Analyses

| Endpoint/ Parameter/ Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Populations | | | |
| Subject Populations | Υ | | |
| Subject Disposition | | | |
| Subject Disposition | Υ | | |
| Reasons for Screen Failure/Run-in Failures | Υ | | Y |
| Subjects by Country and Centre | Υ | | |
| Reasons for Subject Withdrawal | Υ | | Υ |
| Subjects for Whom the Treatment Blind was Broken | | | Y |
| Planned and Actual Treatments | | | Υ |
| Subjects Attending Each Clinic Visit | Υ | | |
| Subjects Withdrawals over Time | | Υ | |
| Protocol Deviations | | | |
| Subjects with Inclusion/ Exclusion/Randomisation Criteria | V | | <b>V</b> [1] |
| Deviations | Υ | | <b>Y</b> [1] |
| Important Protocol Deviations | Υ | | Υ[1] |
| All Protocol Deviations | | | Υ |
| Exclusions from the Per protocol Population | Υ | | |
| Demography and Baseline Characteristics | | | |
| Demographics Characteristics | Υ | | Υ |
| Race and Racial Combinations | Υ | | <b>Y</b> [2] |
| Race and Racial Combination Details | Υ | | |
| Medical Condition | | | |
| Medical Conditions (Current/Past) | Υ | | Υ |
| Past Cholecystectomies | Υ | | Υ |
| Family History of Cardiovascular Risk Factors | Υ | | Υ |
| COPD History | Υ | | Y |
| COPD Exacerbation | Υ | | Y |
| Smoking History and Status | Υ | | Υ |
| Lung Function Test at Screening | Υ | | Υ |
| GOLD Stage and Reversibility/Responsiveness | Υ | | Υ |
| Scores for Modified Medical Research Council dyspnoea | Y | | Y |
| Concomitant Medication | | , | |

| Endpoint/ Parameter/ Display Type | Data | Displays Gene | rated |
|---|---|---|---|
| | Table | Figure | Listing |
| COPD medications not given for an exacerbation taken pre-treatment | Y | | |
| COPD medications not given for an exacerbation taken on-treatment | Y | | |
| COPD medications not given for an exacerbation taken post-treatment | Y | | |
| Medications given for an exacerbation taken pre-treatment | Υ | | |
| Medications given for an exacerbation taken on-treatment | Y | | |
| Medications given for an exacerbation taken post- | Υ | | |
| treatment | • | | |
| Non-COPD medications taken pre-treatment | Υ | | |
| Non-COPD medications taken on-treatment | Υ | | |
| Non-COPD medications taken post-treatment | Υ | | |
| Relationship between ATC Level 1, Ingredient and | | | Υ |
| Verbatim Text | | | Ī |
| COPD medications | | | Υ |
| Non-COPD medications | | | Υ |
| Treatment Compliance | | | |
| Treatment compliance | Y | | Υ |

- Y = Yes display generated.
- All summaries tables will be presented by treatment group and overall.
- COPD History and COPD Exacerbation will be listed together.
- Screening lung function data, GOLD stage, reversibility to salbutamol and reversibility to salbutamol and ipratropium will be listed together.
- COPD and non-COPD medications will be listed separately. The COPD medications listing will indicate whether
  each medication was taken for an exacerbation. Both listings will indicate in which study phases each medication
  was taken (pre-treatment, ontreatment and/or post-treatment).
- [1] Flag shall be provided to identify if the subject is excluded from PP Population or excluded from PP population analysis.
- [2] Listing of race.

#### 7. PRIMARY STATISTICAL ANALYSES

#### 7.1. Primary Efficacy Analyses

#### 7.1.1. Overview of Planned Primary Efficacy Analyses

The primary efficacy analyses will be based on the Modified Intent-To-Treat population, for the analysis on all countries overall and on China Modified Intent-To-Treat population for the analysis on China subgroup alone, unless otherwise specified.

Table 3 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 14: List of Data Displays. All the planned primary efficacy analyses will be done on all countries overall, and China subgroup alone (with the exception of those displays specified by country).

Table 3 Overview of Planned Efficacy Analyses

| Endpoints | | | | Absolu | te | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats<br>Analysis | | Summary | | Indivi | Individual | | Stats Analysis | | | mary | Inc | Individual | |
| | Т | F | L | Т | F | F | L | Т | F | Г | Т | F | F | L |
| <b>Primary Efficacy Analys</b> | es | | | | | | | | | | | | | |
| Baseline FEV <sub>1</sub> | | | | <b>Y</b> [1] | | | Υ | | | | | | | |
| Trough FEV₁ on Day<br>169 | <b>Y</b> [1] | | | <b>Y</b> [1] | | | Y | <b>Y</b> [1 | Y | | <b>Y</b> [1] | Y | | Y |
| Trough FEV₁ on Day<br>169 (Using LOCF) | Υ | | | Y | | | | Υ | | | Y | | | |
| Trough FEV1 at other time points | Υ | | | Y | | | Y | Υ | Υ | | Y | | | Y |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- All the tables will be presented by treatment group.
- [1]: Will be repeated for PP population.

#### 7.1.2. Planned Primary Efficacy Statistical Analyses

#### **Primary Statistical Analyses**

#### Endpoint(s)

Change from baseline in trough FEV1

#### **Model Specification**

- Mixed Models Repeated Measures (MMRM) model.
- While missing data are not explicitly imputed in the primary MMRM analyses, there is an
  underlying assumption that the data are missing at random. All available scheduled
  postbaseline assessments will be utilized and via modeling of the within-subject correlation
  structure, the derived treatment differences will be adjusted to account for missing data.
- The MMRM analysis for trough FEV1 will include on-treatment FEV1 measurements at Days 2, 28, 56, 84, 112, 168 and 169.
- Terms fitted the model:

Response :trough FEV1 on each day or Change from baseline in

trough FEV1 on each Day

Categorical :Treatment, Smoking Status (screening), Country [1],

Day

Continuous :Baseline FEV1

Interaction : baseline\*Day, treatment\*Day

Repeated : Day (nominal)

- The model will be fit with an unstructured variance-covariance matrix.
- The Kenward and Roger method (KR) for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used. In the event the model fails to run using the KR method, then the residual method will be used instead.
- Baseline is defined in Section 10.5.2.1
- Two models will be fitted; one with trough FEV1 on each Day and one with Change from baseline in trough FEV1 on each Day.

#### **Model Checking & Diagnostics**

• Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### Model Results Presentation

- Least-square (LS) means and LS mean change from baseline values for each treatment group will be presented with their associated standard errors.
- Estimated treatment differences along with corresponding 95 % confidence intervals (CIs) and p-values for Days 2, 28, 56, 84,112, 168 and 169 will be presented for the treatment comparisons
- The LS means from the model for change from baseline in trough FEV1 for each treatment on Days 2, 28, 56, 84, 112, 168 and 169, along with the corresponding 95 % CIs, will be plotted.
- The LS mean treatment differences, along with the corresponding 95 % CIs, for change from baseline in trough FEV1 on Days 2, 28, 56, 84, 112, 168 and 169 will be plotted for active treatment group versus placebo.
- The type III tests of fixed effects and the covariance parameter estimates from the model will

#### **Primary Statistical Analyses**

be presented in two tables in the statistical appendix.

#### Example SAS Code

proc mixed data=dsetin;

class trtcd visit subjid smk country[1];

model endpoint=trtcd baseline smk country<sup>[1]</sup> day day\*baseline day\*trtcd / ddfm =kr; repeated visit / subject=subjid type=un:

Ismeans trtcd\*visit / cl diff e om=OMdset at (baseline)=(&blm.);

ods output Ismeans=Ismeans;

ods output diffs=diffs;

run;

[where OMdset is a dataset with a row for every subject-visit combination that contains all of the covariates and blm is a macro variable containing the mean baseline for the subjects used in the analysis. This is used to derive the LS means using coefficients which are based on the subjects used in the analysis.]

Note: [1]: In China subgroup analysis, Country will be removed.

#### Sensitivity and Supportive Statistical Analyses

- The summaries, figures and analysis detailed in Section 7.1.1 (Overview of Planned Efficacy Analyses) and above primary statistical analyses, except for the summary figures (box plot and empirical distribution function plot, details please refer to Appendix 14), will be repeated for the PP population for the analysis on all countries overall and on China PP population for the analysis on China subgroup alone as the supportive analysis of primary efficacy analyses.
- An assessment of whether the effect of treatment on trough FEV1 is modified by smoking status at screening, country [1] or baseline will be made by fitting separate repeated measures models, identical to the model described in the above primary statistical analyses, but also including additional terms for the treatment by smoking status interaction, treatment by country (for the all countries analysis only) interaction and treatment by baseline interaction respectively.
- Additionally, an assessment will be made of whether the effect of treatment on trough FEV1 is modified by the following factors,

ICS use at screening.

Reversibility to salbutamol at screening.

Post-salbutamol percent predicted FEV1 at screening

This will be made by fitting separate repeated measures models, identical to the model described in Primary Statistical Analyses of Section 7.1.2 but also including additional terms for the factor and the factor by treatment interaction.

- If any interaction from these analyses is significant at the 10 % level, further investigation and characterisation of the interaction will be undertaken.
- The interaction p-values from these analyses will be included in the statistical appendix.

Note: [1]: In China subgroup analysis, Country will be removed.

### 7.1.3. Planned Missing Data Sensitivity Statistical Analyses for Trough FEV1

Missing Trough FEV1 on Day 169 will be imputed using LOCF. This only include post-baseline measurements at on-treatment scheduled clinic visits.

#### **Sensitivity Statistical Analyses – LOCF**

#### Endpoint(s)

• Change from baseline in trough FEV1 on Day 169

#### **Model Specification**

- Analysis of Covariance (ANCOVA) model using LOCF
- Terms in the model:
  - **Response**: trough FEV1 or change from baseline in trough FEV1 on Day 169.
  - Categorical: treatment group, smoking status (screening), country<sup>[1]</sup>
  - **Continuous**: baseline FEV1
- Baseline is defined in Section 10.5.2.1
- Two models will be fitted; one with trough FEV1 on Day 169 and one with Change from baseline in trough FEV1 on Day 169.

#### **Model Results Presentation**

- Least-square (LS) means and LS mean change from baseline values for treatment group will be presented with their associated standard errors.
- The estimated treatment difference along with corresponding standard error, 95% CI and p-value will be presented.

#### **Example SAS Code**

```
proc mixed data=dsetin;
class trtcd smk country<sup>[I]</sup>;
model endpoint=trtcd baseline smk country<sup>[I]</sup> / ddfm =kr;
lsmeans trtcd / cl diff e;
ods output lsmeans=lsmeans;
ods output diffs=diffs;
run;
```

Note: [1]: In China subgroup analysis, Country will be removed.

#### 7.2. Secondary Efficacy Analyses

#### 7.2.1. Overview of Planned Secondary Efficacy Analyses

The secondary efficacy analyses will be based on the Modified Intent-To-Treat population, for the analysis on all countries overall and on China Modified Intent-To-Treat population for the analysis on China subgroup alone, unless otherwise specified.

Table 4 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 14: List of Data Displays. All the planned secondary efficacy analyses will be done on all countries overall, and China subgroup alone (with the exception of those displays specified by country).

#### Table 4 Overview of Planned Efficacy Analyses

| Endpoint | | | | Absolu | ıte | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sumr | nary | Individual | | Stats Analysis | | | Summary | | Individual | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| 0-6 h Weighted Mean | Υ | | | Υ | | | Υ | Υ | | | Υ | | | Υ |
| FEV1 on Day 1 | | | | | | | | | | | | | | |
| Baseline Dyspnea | | | | Υ | | | Υ | | | | | | | |
| Index (BDI) | | | | | | | | | | | | | | |
| Transition Dyspnea | Υ | Υ | | Υ | | | Υ | | | | | | | |
| Index (TDI) | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- All the tables will be presented by treatment group.

#### 7.2.2. Planned Secondary Efficacy Statistical Analyses

#### 7.2.2.1. 0-6 h Weighted Mean FEV1 on Day 1

#### Statistical Analyses

#### Endpoint(s)

0-6 h Weighted Mean FEV1

#### **Model Specification**

- ANCOVA Model
- The absolute and change from baseline value of 0-6 h weighted mean FEV1 on Day 1 will be analysed.
- Terms fitted in the ANCOVA model will be include:

Response :Absolute value or change from baseline value of 0-

6 h weighted mean FEV1 on Day 1

Categorical :Treatment, Smoking Status (Screening), Country[1]

Continuous :Baseline FEV1

- Baseline is defined in Section 10.5.2.1
- Two models will be fitted; one with a response variable of change from baseline and one with the response variable as absolute value.

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- LS mean and LS mean change from baseline values for each treatment group will be presented with their associated standard errors.
- Estimated treatment differences along with corresponding 95 % CIs and p-values for Day 1 will be presented for the treatment comparisons.

#### Example SAS Code

proc mixed data=dsetin;

#### **Statistical Analyses**

class trtcd subjid smk country[1];

model endpoint=trtcd baseline smk country[1] / ddfm =kr;

Ismeans trtcd / cl diff e om;

ods output Ismeans=Ismeans;

ods output diffs=diffs;

run;

Note: [1]: In China subgroup analysis. Country will be removed.

#### 7.2.2.2. TDI

#### **Statistical Analyses**

#### Endpoint(s)

TDI

#### **Model Specification**

MMRM

The model will use all available TDI focal scores recorded on Days 28, 84 and 168.

Terms fitted in the model will be include:

Response : TDI focal scores on each day

Categorical :Treatment, Smoking Status (screening), Country[1],

Day

Continuous :BDI focal score

Interaction : BDI focal score \*Day, treatment\*Day

Repeated : Day (nominal)

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- LS means values for each treatment group will be presented with their associated standard errors.
- Estimated treatment differences along with corresponding 95 % CIs and p-values for Days 28, 84 and 168 will be presented for the treatment comparisons.
- The LS means from the model for TDI focal score for Days 28, 84 and 168, along with the corresponding 95 % CIs, will be plotted
  - ✓ The LS mean treatment differences, along with the corresponding 95 % Cls for Days 28, 84 and 168 will be plotted for active treatment group versus placebo

#### **Example SAS Code**

Similar like the code in Section 7.1.2.

#### 7.3. Other Efficacy Analyses

#### 7.3.1. Overview of Planned Other Efficacy Analyses

Other efficacy analyses will be based on the Modified Intent-To-Treat population, for the analysis on all countries overall and on China Modified Intent-To-Treat population for the analysis on China subgroup alone, unless otherwise specified.

Table 5 provides an overview of the planned other efficacy analyses, with further details of data displays being presented in Appendix 14: List of Data Displays. All the planned study population analyses will be done on all countries overall, and China subgroup alone (with the exception of those displays specified by country).

Table 5 Overview of Planned Other Efficacy Analyses

| Endpoint | | | | Absolu | ıte | | | С | hange | from | Basel | ine | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sumr | nary | Indiv | idual | Sta | ats Ana | lysis | Summary | | Individual | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Time to Onset (an | Υ | Υ | | Υ | | | Υ | | | | | | | |
| increase of 100mL in | | | | | | | | | | | | | | |
| FEV1 above baseline) | | | | | | | | | | | | | | |
| during 0-6 h post-dose | | | | | | | | | | | | | | |
| on Day 1 | | | | | | | | | | | | | | |
| Proportion Achieving | Υ | | | Υ | | | Υ | | | | | | | |
| Increase in FEV1 of | | | | | | | | | | | | | | |
| ≥12 % and ≥200 mL | | | | | | | | | | | | | | |
| above Baseline at any | | | | | | | | | | | | | | |
| Time During 0-6 h | | | | | | | | | | | | | | |
| Post-dose on Day 1 Proportion Achieving | Υ | | | Υ | | | Υ | | | | | | | |
| Increase of ≥100 mL | ı | | | ı | | | ı | | | | | | | |
| above Baseline in | | | | | | | | | | | | | | |
| Trough FEV1 | | | | | | | | | | | | | | |
| Serial FEV1 | Υ | Υ | | Υ | | | Υ | Υ | Υ | | Υ | | | |
| Trough FVC | Y | ' | | Y | | | Y | Y | Y | | Y | | | |
| Serial FVC | Y | Υ | | Y | | | Y | Y | Y | | Y | | | |
| Rescue Salbutamol | | | | Y | | | Y | • | | | Y | | | |
| Use (Percentage of | | | | • | | | | | | | | | | |
| Rescue-Free Days)[1] | | | | | | | | | | | | | | |
| Rescue Salbutamol | Υ | | | Υ | | | Υ | Υ | | | Υ | | | Υ |
| Use (mean | | | | | | | | | | | | | | |
| puffs/days)[1] | | | | | | | | | | | | | | |
| Proportion of | Υ | | | Υ | | | Υ | | | | | | | |
| Responders According | | | | | | | | | | | | | | |
| to TDI Focal Score[2] | | | | | | | | | | | | | | |
| Time to First COPD | Υ | Υ | | Υ | | | Υ | | | | | | | |
| Exacerbation | | | | | | | | | | | | | | |
| On-Treatment COPD | | | | Υ | | | | | | | | | | |
| Exacerbations <sup>[3]</sup> | | | | | | | | | | | | | | |
| Post-Treatment COPD | | | | Υ | | | | | | | | | | |
| Exacerbations <sup>[3]</sup> | | | | | | | | | | | | | | |

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- All the tables will be presented by treatment group.
- [1]: Absolute summary will be done on each at baseline, during each four weeks of treatment and over the entire 24-week treatment period. The change from baseline values will also be summarised by treatment, for each four weeks of treatment and the entire 24-week treatment period.
- [2]: A responder to TDI will be defined as a subject with TDI score of 1 unit or more
- [3]: The number and percentage of subjects reporting 0, 1, 2 or >2 on-treatment COPD exacerbations and the total number of exacerbations will be presented by treatment group. The number and percentage of exacerbations with each outcome category, the number and percentage of exacerbations leading to withdrawal and the number and percentage of exacerbations treated by oral/systemic corticosteroids, antibiotics, or which resulted in a visit to the emergency room or hospitalisation will also be presented. In addition, the exacerbation duration will be summarised.

#### 7.3.2. Planned Other Efficacy Statistical Analyses

#### 7.3.2.1. Time to Onset and Time to First COPD Exacerbation

#### **Statistical Analyses**

#### Endpoint(s)

- Time to Onset (an increase of 100mL in FEV1 above baseline) during 0-6 h post-dose on Day
- Time to First COPD Exacerbation

#### Model Specification

- Cox's proportional hazards model
- Terms in the model:

Dependent variable: Time to Onset or time to first COPD exacerbation Categorical: treatment group, smoking status (screening), and Country<sup>[1]</sup>.

• Use the 'exact' method for handling ties. (If the analysis will not run using the 'exact' method, then the 'Efron' method for handling ties will be used instead.)

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Hazard ratios for each of the treatment comparisons with associated 95 % CIs and p-values, will be presented.
- Kaplan-Meier survivor functions of the proportion of subjects with onset over time will be
  obtained for each treatment group separately and will be plotted on the same figure.
- The median time to onset on Day 1 (taken from the Kaplan Meier analysis) will also be presented in the summary table.

#### **Example SAS code**

Cox's proportional hazards model

#### Statistical Analyses

```
proc phreg data=dsetin;
```

model timeto1\*eventflag(0)=treatment smokehis country[1]

/ risklimits ties=exact;

run;

Kaplan-Meier survivor functions

proc lifetest data=wdw outsurv=survest;

time timeto1\*eventflag(0);

strata treatment;

run:

quit;

Note: [1]: In China subgroup analysis, Country will be removed.

#### 7.3.2.2. Proportion Endpoints

#### **Statistical Analyses**

#### Endpoint(s)

- Proportion Achieving Increase in FEV1 of ≥12 % and ≥200 mL above Baseline at any Time During 0-6 h Post-dose on Day 1
- Proportion Achieving Increase of ≥100 mL above Baseline in Trough FEV1
- Proportion of Responders According to TDI Focal Score

#### **Model Specification**

#### **Proportion Endpoints**

- Logistic Regression Model
- At each of Days 2, 28, 56, 84, 112, 168 and 169, the proportion of subjects who achieved an
  increase of 100 mL above baseline in trough FEV1 will be analysed using a separate logistic
  regression model.
- At each visit, the proportion of responders according to TDI focal score will be analysed using a separate logistic regression model.
- Terms in the model:

Dependent Variable : Proportion

Categorical :Treatment, Smoking Status (screening), Country[1]

Continuous :Baseline FEV1 or BDI

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

• For each treatment comparison, the odds ratio, 95 % CI and p-value will be presented.

#### **Example SAS code**

proc logistic data=fevaanal descending;

class treatment (ref='1') smokehis country[1] / param=ref;

model respond=treatment base smokehis country[1] / clodds=wald expb;

ods output logistic.oddsratios=odds1

(where=(index(effect, 'TREATMENT')>0

# or index(effect,'treatment')>0)); ods output logistic.parameterestimates=pval1 (keep=probchisq variable classval0 where=(variable in ('TREATMENT','treatment'))); run;

Note: [1]: In China subgroup analysis, Country will be removed.

#### 7.3.2.3. Serial FEV1/FVC and Trough FVC

#### **Statistical Analyses**

#### Endpoint(s)

- Serial FEV1 (including post dose 15 and 30 min, 1, 3 and 6 h post-dose measurements on Day
   1)
- Trough FVC (including Days 2, 28, 56, 84, 112, 168 and 169)
- Serial FVC (including post dose 15 and 30 min, 1, 3 and 6 h post-dose measurements on Day
   1)

#### Model Specification, Checking, Results Presentation and SAS code

Similar to trough FEV1 in Section 7.1.2

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### 7.3.2.4. Rescue Salbutamol Use (mean puffs/days)

#### **Statistical Analyses**

#### Endpoint(s)

• Rescue Salbutamol Use (mean puffs/days) (absolute and change from baseline value)

#### **Model Specification**

#### ANCOVA model

- The mean number of puffs of rescue medication per day over each four weeks of treatment and the entire 24 week treatment period will be analyzed.
- Terms in model:

Response : Rescue Salbutamol Use (mean puffs/days) (absolute or

change from baseline value)

Fixed Categorical :Treatment, Smoking Status, Country<sup>[1]</sup>

Fixed Continuous Covariates :Baseline
 Baseline is defined in Section 10.6.5 Rescue Use part.

• Two models will be fitted; one with absolute value and one with change from baseline value.

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- LS means and LS mean change from baseline values for each treatment group will be presented with their associated standard errors.
- Estimated treatment differences along with corresponding 95 % CIs and p-values will be presented for the treatment comparisons.

#### Example SAS code

# Statistical Analyses proc mixed data=start; by week; class treatment smokehis country<sup>[1]</sup>; model endpoint=treatment baseline smokehis country<sup>[1]</sup>; Ismeans treatment / cl diff e om; ods output Ismeans=Ismeans; ods output diffs=diffs; run;

Note: [1]: In China subgroup analysis, Country will be removed.

#### 7.4. Health Outcomes Analyses

#### 7.4.1. Overview of Planned Health Outcomes Analyses

Health outcomes analyses will be based on the Modified Intent-To-Treat population, for the analysis on all countries overall and on China Modified Intent-To-Treat population for the analysis on China subgroup alone, unless otherwise specified.

Table 6 provides an overview of the planned health outcomes analyses, with further details of data displays being presented in Appendix 14: List of Data Displays. All the planned study population analyses will be done on all countries overall, and China subgroup alone (with the exception of those displays specified by country).

Table 6 Overview of Planned Health Outcomes Analyses

| Endpoint | | | ı | Absolu | ıte | | | | C | hange | from | Basel | ine | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | lysis | Sum | mary | Indiv | /idual | Sta | ats Ana | lysis | Sum | mary | Individual | |
| | Т | F | L | T | F | F | L | Τ | F | L | T | F | F | L |
| Baseline SGRQ (Total | | | | Υ | | | <b>Y</b> [1] | | | | | | | |
| and each domain) | | | | | | | | | | | | | | |
| SGRQ total score | Υ | | | Υ | | | Υ | Υ | Υ | | Υ | Υ | | Υ |
| SGRQ each domain | | | | Υ | | | Υ | | | | Υ | | | |
| score | | | | | | | | | | | | | | |
| Proportion of | Υ | | | Υ | | | | | | | | | | |
| responders according | | | | | | | | | | | | | | |
| to SGRQ total score | | | | | | | | | | | | | | |
| Baseline COPD | | | | Υ | | | | | | | | | | |
| Assessment Test | | | | | | | | | | | | | | |
| (CAT) score | | | | | | | | | | | | | | |
| CAT score | Υ | | | Υ | <b>Y</b> [2] | | Υ | Υ | | | Υ | | | Υ |
| Proportion of | Υ | | | Υ | | | | | | | | | | |
| Responders according | | | | | | | | | | | | | | |
| to CAT Score | | | | | | | | | | | | | | |
| Healthcare Resource | | | | Υ | | | Υ | | | | | | | |
| Utilisation | | | | | | | | | | | | | | |

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- All the tables will be presented by treatment group.
- [1]: Only total baseline score will be listed.
- [2]: Two scatter plots will be generated:
   Change from baseline CAT score at day 168 vs Change from baseline FEV1 at 168
   Baseline CAT scores versus baseline FEV1

#### 7.4.2. Planned Health Outcomes Statistical Analyses

#### **Primary Statistical Analyses**

#### Endpoint(s)

- SGRQ
- CAT score
- Proportion of responders according to SGRQ total score

#### Model Specification, Checking, Results Presentation and SAS code

#### SGRQ,

#### CAT score

Similar to trough FEV1 in Section 7.1.2

#### Proportion of responders according to SGRQ total score Proportion of Responders according to CAT Score

• Similar to proportion endpoint in Section 7.3.2.2

#### 8. SAFETY ANALYSES

#### 8.1. Adverse Events Analyses

#### 8.1.1. Overview of Planned Adverse Events Analyses

The safety analyses will be based on the Modified Intent-To-Treat population, for the analysis on all countries overall and on China Modified Intent-To-Treat population for the analysis on China subgroup alone, unless otherwise specified.

In case of treatment misallocation, additional outputs for safety analyses may be provided, showing the subjects impacted by misallocation and the treatments they actually received.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays. All the planned study population analyses will be done on all countries overall, and China subgroup alone (with the exception of those displays specified by country).

Table 7 Overview of Planned Adverse Event Analyses

| Endpoint | | Abso | lute |
|---|---|---|---|
| · | Sumi | mary | Individual |
| | Т | F | L |
| Exposure | | | |
| Exposure to Study Treatment | Υ | | Υ |
| Adverse Events (AEs) | | | |
| Overview of AE incidence | | | |
| All AEs by SOC | Υ | | Υ |
| Common AEs by Overall Frequency | Υ | Υ | |
| All Drug-Related AEs by SOC | Υ | | |
| Subject Numbers for Individual AEs | | | Υ |
| Relationship Between AE SOCs, PT & Verbatim Text | | | Υ |
| On-Treatment AEs by SOC | Υ | | |
| Post-Treatment AEs by SOC | Υ | | |
| On-Treatment AEs experienced by 3% (after rounding) or more of subjects in | Υ | | |
| any treatment group | | | |
| Common On-Treatment non-serious AEs[1] | Υ | | |
| On-treatment Drug-Related AE's | Υ | | |
| On-treatment Non-Serious Drug Related Adverse Events | Υ | | |
| All AEs | | | Υ |
| Serious and Other Significant AEs | | | |
| Fatal SAEs[1] | Υ | | Y |
| Non-Fatal SAEs | Υ | | Υ |
| Pre-treatment fatal SAEs | Υ | | |
| Pre-treatment non-fatal SAEs | Υ | | Υ |
| On-treatment non-fatal SAEs | Υ | | Υ |
| Post-treatment Non-fatal SAEs | Υ | | Υ |
| SAEs by SOC | Υ | | |
| Drug related serious AE | Υ | | |

| Endpoint | Absolute | | |
|---|---|---|---|
| | Sumr | nary | Individual |
| | Τ | F | L |
| Drug related SAEs by SOC | | | Υ |
| Pre-treatment AEs leading to withdrawal from the study | Υ | | Υ |
| On-treatment AEs leading to permanent discontinuation of study treatment or | Υ | | Υ |
| withdrawal from the study | | | |
| On-Treatment AE of Special Interest | Υ | | Υ |
| Fatal SAE of Special Interest | Υ | | |
| On-treatment Non-Fatal SAE of Special Interest | Υ | | |
| Drug Related Fatal SAEs | Υ | | |
| On-treatment Non-Fatal Drug Related SAEs | Υ | | |
| Reasons for potential ELLIPTA malfunctions | | | Y |

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- All the tables will be presented by treatment group.
  - [1]: A cut-off of 3% for 'common' will be used, but for this purpose it should be applied without rounding, i.e. an event experienced by 2.8% subjects should not be included. This table also needs a 'number of subjects with any event' row which only counts subjects experiencing any event in the body of the table.

#### 8.2. Clinical Laboratory Analyses

#### 8.2.1. Overview of Planned Clinical Laboratory Analyses

The safety analyses will be based on the Modified Intent-To-Treat population, for the analysis on all countries overall and on China Modified Intent-To-Treat population for the analysis on China subgroup alone, unless otherwise specified.

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays. All the planned study population analyses will be done on all countries overall, and China subgroup alone (with the exception of those displays specified by country).

Table 8 Overview of Planned Clinical Laboratory Analyses

| Endpoint | | Abs | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sumn | nary | Indiv | idual | Summary | | y Individua | |
| | T | F | F | L | Т | F | F | L |
| Chemistry | | | | | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry | Υ | | | | Υ | | | |
| Clinical Chemistry values outside the normal range | Υ | | | Υ | | | | |
| Clinical Chemistry change from baseline value relative to | Υ | | | | | | | |
| the normal range | | | | | | | | |
| Clinical Chemistry maximum post-baseline value | | Υ | | | | Υ | | |
| Clinical Chemistry minimum post-baseline value | | Υ | | | | Υ | | |
| Hematology | | | | | | | | |
| Hematology | Y | | | | Υ | | | |
| Hematology values outside the normal range | Y | | | Υ | | | | |

| Endpoint | Absolute | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Summ | ary | Individual | | Summary | | Individual | |
| | Т | F | F | L | T | F | F | L |
| Hematology change from baseline value relative to the | Υ | | | | | | | |
| normal range | | | | | | | | |
| Hematology maximum post-baseline value | | Υ | | | | Υ | | |
| Hematology minimum post-baseline value | | Υ | | | | Υ | | |
| Urinalysis | | | | | | | | |
| Urinalysis data | Υ | | | Υ | | | | |
| Hepatobiliary (Liver) | | | | | | | | |
| Liver Event | | | | Y | | | | |

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.3. Other Safety Analyses

#### 8.3.1. Overview of Planned Other Safety Analyses

The safety analyses will be based on the Modified Intent-To-Treat population, for the analysis on all countries overall and on China Modified Intent-To-Treat population for the analysis on China subgroup alone, unless otherwise specified.

Table 9 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays. All the planned study population analyses will be done on all countries overall, and China subgroup alone (with the exception of those displays specified by country).

Table 9 Overview of Planned Other Safety Analyses

| Endpoint | Absolute | | | | | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| - | Stats Analysis | | | Summary Individual | | | Stats Analysis | | | Summary | | Individual | | |
| | Т | F | Г | Т | F | F | L | Т | F | L | Т | F | F | L |
| Vital Signs | Vital Signs | | | | | | | | | | | | | |
| Pulse rate | Υ | Υ | | Υ | | | Υ | Υ | | | Υ | | | Υ |
| Systolic | Υ | Υ | | Υ | | | Υ | Υ | | | Υ | | | Υ |
| Diastolic blood | Υ | Υ | | Υ | | | Υ | Υ | | | Υ | | | Υ |
| pressure | | | | | | | | | | | | | | |
| 12-Lead ECG | | | | | | | | | | | | | | |
| QTc(F) | Υ | Υ | | Υ | Υ | | | Υ | | | Υ | Υ | | |
| QTc(B) | | | | Υ | | | | | | | Υ | | | |
| PR interval | Υ | Υ | | Υ | | | | Υ | | | Υ | | | |
| Heart Rate | Υ | Υ | | Υ | | | | Υ | | | Υ | | | |
| ECG interpretation | | | | Υ | | | | | | | | | | |
| ECG abnormalities | | | | Υ | | | Υ | | | | | | | |

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- All the tables will be presented by treatment group.

#### 8.3.2. Planned Safety Statistical Analyses

#### **Primary Statistical Analyses**

#### Endpoint(s)

- Pulse rate
- Systolic
- Diastolic blood pressure
- QTc(F)
- PR interval
- Heart Rate

#### **Model Specification**

- ANCOVA model
- The absolute and change from baseline value of each endpoint will be statistically analysed at each scheduled time point after the start of treatment separately.
- Terms fitted in the ANCOVA model will be include:

Response : Absolute value or change from baseline value at

each scheduled time point.

Fixed Categorical :Treatment, Smoking Status(Screening), Country[1]

Fixed Continuous Covariates :Baseline

- Baseline is defined in Section 10.5.2.1.
- Two models will be fitted; one with a response variable of change from baseline and one with the response variable as absolute value.

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Treatment group LS mean values and LS mean change from baseline values with associated standard errors will be presented for each scheduled on-treatment time point for each endpoint.
- LS mean treatment differences for comparisons will be presented with associated 95 % Cls.
- LS mean change from baseline and associated 95 % CIs for pre-dose values at each scheduled time point by treatment group will be presented graphically.

#### **Example SAS Code**

Similar to the code in Section 7.2.2.2

Note: [1]: In China subgroup analysis, Country will be removed.

#### 9. REFERENCES

CPMP/EWP/562/98. Points to Consider on Clinical Investigation of Medicinal Products in the Chronic Treatment of Patients with Chronic Obstructive Pulmonary Disease (COPD). 19 May 1999

GlaxoSmithKline Document Number 2013N159587\_03 Study ID AC4117410. A 24-week randomised, double-blind and placebo-controlled study to evaluate the efficacy and safety of 62.5 mcg Umeclidinium Inhalatin Powder delivered once-daily via a Novel Dry Powder Inhaler in subjects with Chronic Obstructive Pulmonary Disease Effective Date: 11-NOV-2015.

Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2011. Available from: http://www.goldcopd.org/.

ICH E1A. The Extent of Population Exposure to Assess Clinical Safety: For Drugs intended for Long Term Treatment of Non-Life Threatening Conditions.

Siddiqui O, Hung HMJ, O'Neill, R. MMRM vs. LOCF: A Comprehensive Comparison Based on Simulation Study and 25 NDA Datasets J Biopharm Stat 2009; 19:227-46.

St. George's Respiratory Questionnaire Manual, Version 2.3, 2009.

Witek TJ, Jr., Mahler DA. Minimal important difference of the transition dyspnoea index in a multinational clinical trial. Eur Respir J 2003; 21:267-272.

#### 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Assessment Windows |
| Section 10.4 | Appendix 4: Treatment States & Phases |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 10.9 | Appendix 9: Multicentre Studies |
| Section 10.10 | Appendix 10: Examination of Covariates and Subgroups |
| Section 10.11 | Appendix 11: Multiple Comparisons and Multiplicity |
| Section 10.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 10.13 | Appendix 13: Abbreviations & Trade Marks |
| Section 10.14 | Appendix 14: List of Data Displays |
| Section 10.15 | Appendix 15: Example Mock Shells for Data Displays |

## 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Protocol deviations identified in this section are those considered to affect the primary outcome of the study. All decisions on whether to exclude a subject or a subject's data from analysis will be made prior to breaking the blind, with the exception of subjects receiving incorrect treatment container. If, after breaking the blind, the container was found to have contained the correct randomised treatment, no data will be excluded from analyses.

#### 10.1.1. Exclusion of Data from Modified Intent-to-treat Analyses

In general, all data recorded for subjects who were randomised and received at least one dose of study medication will be included in Modified ITT analyses. The following deviations will result in exclusion of data from Modified ITT analyses:

If a 23 h or 24 h post-dose FEV1 or FVC assessment is actually performed after the following day's dose, the value will be excluded from Modified ITT analyses.

If a 15 or 30 min, 1, 3, or 6 h FEV1 or FVC assessment is actually performed before dosing, the value will be excluded from Modified ITT analyses.

Derived endpoints will be calculated from remaining assessment values. Exclusion of a value from Modified ITT analyses does not necessarily mean the subject will not have a value for the derived endpoints.

#### 10.1.2. Exclusions of Data from Per Protocol Analyses

Subjects with full protocol deviations identified below will be excluded from the PP population. Subjects with partial protocol deviations will generally be included in the PP population but have data excluded from PP analyses from the time of the deviation onwards. The exception to this is a partial deviation which occurred prior to the start of treatment – in this case the subject will be excluded from the PP population. Subjects with time-point specific deviations will have only the affected data excluded from PP analyses.

#### 10.1.2.1 Inclusion/exclusion/randomisation Criteria Deviations

Failure of criteria will be considered a full protocol deviations as detailed in Table 10:

Table 10 Inclusion/exclusion/randomisation criteria deviations considered to affect the primary outcome

| Reason for exclusion | Full protocol deviation considered to affect primary outcome |
|---|---|
| Inclusion criterion | |
| Type of subject | No |
| Informed consent | No |
| Age | Yes |
| Gender | No |
| COPD History | Yes |
| Tobacco Use and Smoking history | Yes |
| Severity of disease | Yes |
| Dyspnoea (mMRC) | Yes |
| Exclusion criterion | |
| Pregnancy | No |
| Asthma | Yes |
| Other respiratory disorders | Yes |
| Other diseases/abnormalities | No |
| Chest X-ray | Yes |
| Contraindications | No |
| Hospitalisation | Yes |
| Lung resection | Yes |
| 12-lead ECG | No |
| Screening labs | No |
| Medication prior to spirometry | Yes |
| Medication prior to screening | Yes |
| Oxygen | Yes |
| Nebulised therapy | No |
| Pulmonary rehabilitation | Yes |
| Drug or alcohol abuse | No |
| Affiliation with investigator site | No |
| Compliance | No |
| Randomisation criterion | |
| Pre-dose 12-Lead ECG at Visit 2 | No |
| COPD exacerbation | Yes |
| ICS | Yes |
| Prohibited Medications | Yes |

#### 10.1.3. Programmed Checks to Identify Non-medication Deviations

The data checks identified in Table 11 will be performed to further identify protocol deviations.
Table 11
 Programmed non-medication checks

| Reason for exclusion | Check performed | Deviation Type |
|---|---|---|
| Age | (visit date – date of birth) < 40 at prescreening | Full |
| Smoking history | number of pack-years < 10 at screening <sup>[1]</sup> or only use a pipe and/or cigar | Full |
| Severity of disease: FEV1/FVC | Pre-salbutamol or Post-salbutamol FEV₁/FVC ≥0.7 or any one missing at screening | Full |
| Severity of disease: % predicted | Pre-salbutamol or Post-salbutamol FEVPDPC > 70% or any one missing at screening | Full |
| Dyspnea (mMRC) | mMRC < 2 at screening or missing | Full |
| COPD exacerbation during run-in | Exacerbation onset date between dates of screening and start of treatment | Full |
| Compliance with treatment | Overall compliance < 80 % or > 120 % or missing | Full |
| Incorrect treatment | At any point | Partial; data excluded from start of incorrect treatment onwards |
| Blind broken <sup>[3]</sup> | At any point | Partial; data excluded from date of breaking of blind |
| COPD exacerbation during treatment and not withdrawn | Exacerbation onset date between treatment start and stop date +1 with measurement of primary efficacy endpoint after onset date <sup>[2]</sup> | Partial; data excluded from date of onset onwards |
| Meet other withdrawn criteria defined in the protocol but not withdrawn | Manual Review | Partial; data excluded from date of PD happened. |
| Trough FEV1 outside window | 23 h or 24 h FEV1 assessment outside window of 22.5-24.5h after previous day's dose | Time-point specific |

#### Note:

- 1. Pipe and/or cigar use cannot be used to calculate pack-year history.
- 2. Subject experiences an exacerbation during the treatment period requiring the use of any systemic or oral corticosteroids with prescribed or non-prescribed (self-administered) antibiotics, and/or requiring emergency treatment or hospitalisation. If subjects used either prescribed or non-prescribed (self-administered) antibiotics only for the treatment of exacerbation, they were permitted to remain in the study under Pl's discretion according to the study protocol therefore the use of only antibiotics will not be defined as a protocol deviation.
- 3. Subjects whose blind was broken by someone external to GSK (i.e. site staff).

#### 10.1.4. **Programmed Checks to Identify Medication Deviations**

Medications will be classified into Respiratory Medication Class (RMC) as identified in concomitant medications part of Section 10.6.3.

Following agreement of the correct classification, medications taken prior to or ontreatment (i.e. medication start date on or before treatment stop date) in the intervals identified in Table 12 will be reviewed to identify data which should be excluded from analysis. If the disallowed medication started within the specified window prior to Visit 2 the deviation will be considered full and the subject will be excluded from the PP population. Otherwise the deviation will be considered partial and the subject's data will be excluded from PP analyses from the start of the disallowed medication onwards.

Table 12 **Programmed medication checks** 

| RMC | Disallowed rule |
|---|---|
| Depot corticosteroids | Started on-treatment; stopped after 12 weeks prior to V1 |
| Systemic, oral, parenteral and intra-articular corticosteroids | Started on-treatment; stopped after 4 weeks prior to V1. |
| Antibiotics <sup>1</sup> | Stopped after 4 weeks prior to V1, and reason is LRTI <sup>1</sup> |
| ICS <sup>2</sup> | Started on-treatment; stopped after 30 days prior to V1 <sup>2</sup> |
| PDE4 inhibitors | Started on-treatment; stopped after 14 days prior to V1 |
| Long-acting anticholinergics | Started on-treatment; stopped after 7 days prior to V1 |
| Xanthines | Started on-treatment; stopped after 12 hours prior to each visit |
| Leukotriene receptor antagonists | Started on-treatment; stopped after 2 days prior to V1 |
| Oral beta-2 agonists – long acting <sup>3</sup> | Started on-treatment; stopped after 2 days prior to V1 |
| Oral beta-2 agonists - short-acting | Started on-treatment; stopped after day of V1 |
| Inhaled beta-2 agonists – long acting <sup>3</sup> | Started on-treatment; stopped after 2 days prior to V1 |
| Nedocromil or sodium cromoglycate | Started on-treatment; stopped after 1 day prior to V1 and route is inhaled |
| Other investigational medication for COPD | Started on-treatment; stopped after 30 days prior to V1 |
| Any investigational medication | 30 days or 5 half lives, whichever is longer |
| Oxygen | Greater than 12 hours a day |
| Herbal medicine for respiratory diseases | Manual Review |

<sup>1.</sup> All antibiotics will be identified; manual review to identify those with reason for administration of LRTI. After v1, antibiotics used for acute infection <=2weeks is permitted.

Started but not as switch from ICS/LABA or not within allowed dose range

Dose>1000 mcg fluticasone propionate or equivalent

Stopped with no change to an alternative steroid in the same dose range within 14 days of stopping Change dose before treatment or change of more than one dose range on the treatment

<sup>2.</sup> All ICS will be identified; manual review to identify ICS:

<sup>3.</sup> The definition of LABA has now changed and split in to three categories which are now:

<sup>&#</sup>x27;Long-acting beta-2 agonist – Group 1';


```
'Long-acting beta-2 agonist – Group 2 (Olodaterol or Indacaterol)'; 'Long-acting beta-2 agonist – Group 3 (Salmeterol and Formoterol)';
```

The final decision on exclusion will be made following manual review and will be documented prior to unblinding.

# 10.2. Appendix 2: Time & Events

# 10.2.1. Protocol Defined Time & Events

| | | Run-in | | | Doub | le-blind to | reatment | period | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Visit<br>0<br>(Pre-<br>Screen) | Screenin<br>g Visit<br>(Visit 1) | Visit<br>2 | Visit<br>3 | Visit<br>4 | Visit<br>5 | Visit<br>6 | Visit<br>7 | Visit<br>8 | Visit<br>9 | Early<br>With-<br>drawal<br>(EW) Visit | Follow-Up<br>(Phone<br>contact) |
| Day | | Day<br>-7 to -14 | Day<br>1 | Day<br>2 | Day<br>28±2 | Day<br>56±4 | Day<br>84±4 | Day<br>112±4 | Day<br>168±4 | Day<br>169<br>(Visit<br>8 +1<br>day) | | 7±2 days after<br>Visit 9 or EW |
| Week | | -1 | 0 | 0 | 4 | 8 | 12 | 16 | 24 | | | |
| Written Informed Consent <sup>1</sup> | x | | | | | | | | | | | |
| Demography/ COPD History | X | | | | | | | | ĵ | | | |
| Medical History | | X | | | | | | | | | Ü | |
| Physical Examination | | X | | | | | | | X | | X | |
| Smoking Status | | X | | | | | | | X | | X | |
| Smoking Cessation Counselling | | X | | | | | | | X | | Х | |
| Chest X-ray <sup>2</sup> | | X | | | | | | | | | - | |
| Inclusion/exclusion criteria | | X | | | | | | | 1 | | Ü . | |
| Randomization criteria | | | X | | | | | | | | 0 | |
| Screening spirometry (including post-<br>bronchodilator testing) <sup>3</sup> | | Х | | | | | | | | | | |
| mMRC questionnaire | | X | | | | | | | | | j i | |
| Register visit in IVSR | х | х | X | X | X | X | X | X | X | X | х | X |
| Diary Card Dispense or<br>Collection/Review | | Х | X | Х | X | X | X | X | X | X | Х | |

| | | Run-in | | | Double-blind treatment period | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Visit<br>0<br>(Pre-<br>Screen) | Screenin<br>g Visit<br>(Visit 1) | Visit<br>2 | Visit<br>3 | Visit<br>4 | Visit<br>5 | Visit<br>6 | Visit<br>7 | Visit<br>8 | Visit<br>9 | Early<br>With-<br>drawal<br>(EW) Visit | Follow-Up<br>(Phone<br>contact) |
| Day | | Day<br>-7 to -14 | Day<br>1 | Day<br>2 | Day<br>28±2 | Day<br>56±4 | Day<br>84±4 | Day<br>112±4 | Day<br>168±4 | Day<br>169<br>(Visit<br>8 +1<br>day) | | 7±2 days after<br>Visit 9 or EW |
| Week | | -1 | 0 | 0 | 4 | 8 | 12 | 16 | 24 | | | |
| Efficacy assessments | 1 | | | | | | | | 1 1 | | | |
| Trough Spirometry <sup>4</sup> | | | | X | X | Х | X | X | X | X | | |
| Serial Spirometry <sup>5</sup> | | | X | | | | | | | | | |
| COPD exacerbation assessment | X | X | Х | X | X | Х | X | X | X | Х | X | X |
| Baseline Dyspnea Index (BDI) | | | X | | | | | | | | | |
| Transition Dyspnea Index (TDI) | | | | | X | | X | | X | | | |
| SGRQ | | | X | | X | | X | v. | X | | | |
| COPD Assessment Test (CAT) | | | Х | | Х | | X | | X | | | |
| Healthcare resource utilization <sup>6</sup> | | | 4 | | | | | | | | <b>—</b> | |
| Safety Assessments | j | | | | | | | | | | | |
| 12-Lead ECG | | X | X7 | | | | χ7 | | X7 | | X | |
| Vital Signs (blood pressure and pulse rate )8 | | X | X | X | X | Х | X | X | X | X | X | |
| Adverse Event /Con-Med Assessment | | X | X | X | X | X | X | X | X | X | X | X |
| Laboratory Assessments | | | | | | | | | | | | |
| Pharmacogenetics sample <sup>9</sup> | | | X | | | | | | | | | |
| Routine urine | | X | | | | | | | X | | X | |
| Urine Pregnancy Test | | X | X | | | | X | | X | | X | X |
| Clinical Laboratory tests <sup>10</sup> | | Χ | | | | | X | | X | | X | |
| Medication | | | | | | | | | | | | |
| COPD and Concurrent Medication<br>Assessment | x | X | X | X | X | Х | X | X | X | Х | X | |

| | | Run-in | Double-blind treatment period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Visit<br>0<br>(Pre-<br>Screen) | Screenin<br>g Visit<br>(Visit 1) | Visit<br>2 | Visit<br>3 | Visit<br>4 | Visit<br>5 | Visit<br>6 | Visit<br>7 | Visit<br>8 | Visit<br>9 | Early<br>With-<br>drawal<br>(EW) Visit | Follow-Up<br>(Phone<br>contact) |
| Day | | Day<br>-7 to -14 | Day<br>1 | Day<br>2 | Day<br>28±2 | Day<br>56±4 | Day<br>84±4 | Day<br>112±4 | Day<br>168±4 | Day<br>169<br>(Visit<br>8 +1<br>day) | | 7±2 days after<br>Visit 9 or EW |
| Week | 1 | -1 | 0 | 0 | 4 | 8 | 12 | 16 | 24 | | | |
| Dispense/collect rescue<br>salbutamol/albuterol | | Х | X | X | X | X | X | X | X | X | X | |
| Dispense double-blind study drug | | | X | | Х | X | X | X | | | | |
| Collect double-blind study drug | | | | | X | X | X | X | X | | X | |
| Assess double-blind study drug compliance | | | | | X | Х | X | Х | X | | Х | |

- 1. Written informed consent must be obtained prior to performing any Visit 1 procedures or initiating any alterations in a subject's medications. Subjects will be assigned a study number at the time the ICF is signed. Visit 0 and Visit 1 may occur on the same day if applicable.
- 2. To be performed only if there is no chest X-ray or CT scan available within 6 months prior to Visit 1
  3. Spirometry to be conducted as follows: pre-bronchodilator testing following by post-albuterol/salbutamol testing, followed by post-ipratropium testing. Post albuterol/salbutamol testing conducted 10 to 30 min after subject self-administration of 4 puffs of albuterol/salbutamol via MDI with a spacer. Subject will then self administer 4 puffs of ipratropium bromide via MDI and spacer, followed by spirometry testing 30 to 60 min later.

- Trough spirometry obtained twice: at 23 and 24 hours after the previous day's morning dose.
   6 hr serial spirometry: Performed post-dose at 15 and 30 min and 1, 3 and 6 hours. At Visit 2 (Day 1), pre-dose measurements will be obtained -30min and -5min pre-dose.
   Healthcare resource utilization will be collected and entered in the e-CRF as required during the study, collection of this data to be aided by the subject documentation in the paper diary of any contact with the doctor or nurse about their lung condition which was unrelated to study participation.
- 7. ECG conducted pre-dose and 10 and 45 minutes post-dose
- Vital signs to be measured pre-dose and 10 and 45 minutes post-dose at visit 2, and measured only pre- dose at other visits (prior to spirometry).
   PGx sample preferably to be obtained at Visit 2 after randomization, but can also be obtained at a subsequent study visit. PGx consent must be obtained prior to sampling.
- 10. Haematology, and clinical chemistry.

## 10.3. Appendix 3: Assessment Windows

Data are generally reported according to the nominal time of clinic visits and assessments as specified in the protocol, and time windows for exclusion will not be defined. For example, if a subject recorded values for the Week 4 visit that were actually made on the 21st day of treatment, they will be presented as Week 4 values in the summary tables.

For the 23 and 24 h post-dose trough FEV1 measurements, a time window of 22.5-24.5 h is allowed for the actual time of an assessment relative to time of dosing. Values falling outside of this window will not be used in the PP analysis of the primary endpoint, but will still be included in all Modified ITT analyses.

## 10.4. Appendix 4: Treatment States and Phases

#### 10.4.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment, unless otherwise specified.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

#### NOTES:

• If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### 10.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

#### 10.4.2.1. Treatment States for Concomitant Medications Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Medication start date < Study Treatment Start Date |
| On-Treatment | Medication start date ≤ Study Treatment Stop Date and Medication stop date≥ Study Treatment Start Date |
| Post-Treatment | Medication stop date > Study Treatment Stop Date |

#### NOTES:

- A medication will be classed in every period of the study in which it was taken.
- For medications with partial start and stop dates or missing start/stop dates, the medication will be classed in every period of the study in which it could have been taken.
- If the study treatment stop date is missing then the medication will be considered to be On-Treatment.
- The answers to the questions "Taken Prior to Study?" and "Ongoing?" which are recorded on the eCRF will also
  be taken into consideration to determine if the medication was started pre-treatment or continued post-treatment.
  In each case, should the answers suggest a different classification than the dates, the medication will be
  summarised in all possible classifications (pre/on/post) in which it could conceivably have been taken.

#### 10.4.2.2. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop +1 |
| Post-Treatment | AE Start Date > Study Treatment Stop Date+1 |
| Onset Time | If Treatment Start Date > AE Onset Date |
| Since 1st Dose | = AE Onset Date - Treatment Start Date |
| (Days) | If Treatment Start Date ≤ AE Onset Date |
| | = AE Onset Date - Treatment Start Date +1 |
| | Missing otherwise. |

| Treatment State | Definition |
|---|---|
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on Inform/CRF OR value is missing. |

#### NOTES:

- If the study treatment stop date is missing then the AE will be considered to be On-Treatment.
- If the AE onset date is missing or partial then the AE will be considered on-treatment unless there is evidence to the contrary (e.g. the month of the onset date is present and is less than the month of the first dose of study treatment).
- AEs reported by subjects who did not receive treatment will be considered pre-treatment.
- Any SAEs for screen failures, run-in failures or subjects who were randomised but did not receive treatment will be classified as pre-treatment SAEs.

#### 10.4.2.3. Treatment States for COPD exacerbation

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Exacerbations Onset Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Exacerbations Onset Date ≤ Study Treatment Stop +1 |
| Post-Treatment | Exacerbations Onset Date > Study Treatment Stop Date+1 |
| Time to first on-<br>treatment<br>exacerbation | = Exacerbation Onset Date of first on-treatment exacerbation - Treatment Start Date +1 Missing otherwise. |
| Duration (Days) | Exacerbation resolution date or date of death – Exacerbation Onset Date + 1 |

#### NOTES:

- If the study treatment stop date is missing then the exacerbation will be considered to be On-Treatment.
- If the exacerbation onset date is missing or partial then the exacerbation will be considered on-treatment unless there is evidence to the contrary (e.g. the month of the onset date is present and is less than the month of the first dose of study treatment).
- Exacerbations reported by subjects who did not receive treatment will be considered pre-treatment.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

#### 10.5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Code | Description | Description | Order [1] |
| Α | UMEC 62.5 mcg | UMEC 62.5 mcg | 2 |
| Р | Placebo | Placebo | 1 |

#### NOTES:

#### 10.5.2. Baseline Definition & Derivations

#### 10.5.2.1. Baseline Definitions

For all endpoints (expect FEV1 and FVC) the baseline value will be the latest pre-dose assessment at schedule visit. Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

The baseline value for FEV1 and FVC is calculated from the values measured 30 min and 5 min pre-dose on Day 1. If the actual time of an assessment is after the time of dosing on Day 1, the value at that assessment will be set to missing prior to calculating baseline. If one of the values is missing then the baseline will be the single remaining value; otherwise the baseline will be the mean of the two values.

| 10.5.2.2. Derivations and Handling of Missing Baseline Data | 10.5.2.2. | Derivations | and Handling of | f Missina | Baseline Data |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = On-treatment Value – Baseline value |
| % Change from Baseline | = 100 x [(On-treatment Value –<br>Baseline value) / Baseline value] |
| Maximum<br>Change from<br>Baseline | = Calculate the change from baseline at each given timepoint and determine the maximum change |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- If either the baseline or on-treatment value is missing then the change from baseline will be set to missing.
- The change from baseline will not be calculated for baseline records or records prior to baseline

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

#### 10.5.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently su | pported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : \arenv\arprod\gsk573719\ac4117410\final |
| QC Spreadsheet | : arenv\arprod\gsk573719\ac4117410\final\qc |
| Analysis Datasets | |
| Analysis datasets will be created according to Integrated Data Standards Library standards. | |
| Generation of RTF Files | |
| RTF files will be generated. | |

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the randomized treatment the subject received unless otherwise stated. However, there may be additional adhoc displays for individual subjects using the actual treatment received.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

 Unscheduled visits will not be included in summary tables except as part of a 'worst case postbaseline' assessment.


AC4117410

| Reporting Standards | |
|---|---|
| <ul> <li>Unscheduled visit</li> </ul> | Unscheduled visits will not be included in figures. |
| All unscheduled | All unscheduled visits will be included in listings. |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. **General**

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

Calculated as the number of days from randomisation date:

- Ref Date = Missing → Study Day = Missing
- Ref Date < Start of treatment date → Study Day = Ref Date Start of treatment date
- Ref Data ≥ Start of treatment date → Study Day = Ref Date (Start of treatment date) + 1

#### **Date of Completion/Withdrawal**

The date of completion/withdrawal will be derived as follows:

- For subjects who complete the last on-treatment study visit, the date of completion/withdrawal will be the date of that visit (Visit 9).
- For subjects who withdraw from the study, the date of completion/withdrawal will be the
  latest of the date of the last attended scheduled clinic visit (excluding follow-up), the date of
  the EW visit (if present) and the last dose date.

## 10.6.2. Study Population

#### **Demographics**

#### Age

- Age will be calculated based on the Pre-screening visit date.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

#### **Smoking Status**

At Screening, subjects who were identified as former smokers but who last smoked within 6 months prior to Screening will be re-classified as current smokers prior to summarizing. Subject listings will include original and re-classified status.

During the study, smoking status will be derived from smoking status at Screening and records of change in smoking status at visits. A subject identified as a current smoker at Screening who stopped smoking during the study will be assessed as a former smoker only at visits which are at least 6 months after the date the subject last smoked. Former smokers who started smoking will be considered current smokers at all visits after the date the subject started smoking.

In order to assess the last time a subject smoked the partial date will be imputed to earliest date within the month or year e.g. If a subject has only remembered the year they last smoked (-----2010) then impute to 01JAN2010. If a subject has remembered the month and year that they last smoked (--SEP2010) then impute to 01SEP2010.

#### **Concomitant Medications**

COPD concomitant medications will be grouped into the following RMCs based on predefined code lists derived from ATC classifications:

```
Short-acting anticholinergic
Short-acting beta-2 agonist
Long-acting anticholinergic
Long-acting beta-2 agonist - Group 1
Long-acting beta-2 agonist - Group 2 (Olodaterol or Indacaterol)
Long-acting beta-2 agonist - Group 3 (Salmeterol and Formoterol)
Xanthine
PDE4 Inhibitors
Corticosteroid - Inhaled
Corticosteroid - Depot
Corticosteroid - Systemic, oral, parenteral and intra-articular
Corticosteroid - Other
Leukotriene Receptor Antagonist
Nedocromil or Cromolyn Sodium
Mucolytics
Cytochrome P450 3A4 Strong Inhibitors
Oxygen
Antiinfectives (antibiotics, antifungals, antivirals, antiseptics)
Other medication given for exacerbation
Other COPD medication
Other
```

COPD concomitant medications that were stopped more than 30 days prior to Screening and non COPD concomitant medications that were stopped prior to Screening will not be presented in any tables or listings.

For reporting purposes, the LABA groups will be combined in the concomitant medication tables.

#### **Treatment Compliance**

The number of doses of study treatment taken by each subject from each inhaler will be calculated from the dose counter start and stop counts for each inhaler used. If a dose counter start count is missing then it will be assumed to be 30. If all dose counter stop counts are non-missing then the percentage compliance will be calculated as:

```
Compliance = \underline{\text{sum of all (dose counter start - dose counter stop)}} \times \underline{100}
(exposure stop date – exposure start date +1)
```

If any dose counter stop is missing then the treatment compliance will be set to missing for that subject.

Overall compliance will be categorised as follows:

```
< 80 \%

\ge 80 \% \text{ to } < 95 \%

\ge 95 \% \text{ to } \le 105 \%

> 105 \% \text{ to } \le 120 \%

> 120 \%.
```

If a subject received a treatment other than the randomised treatment during the study, the compliance will still be calculated using data from all containers received and overall exposure start and stop dates.

# 10.6.3. Safety

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:

   Direction of Exposure in Days Overall Treetment Step Date Overall Treetment
  - Duration of Exposure in Days = Overall Treatment Stop Date Overall Treatment Start

    Date + 1
- If there are any treatment breaks during the study, exposure data will be adjusted accordingly.
- If overall treatment stop date is missing it will be imputed as follows:
  - For subjects who attended a Study Treatment Discontinuation visit, use the date of the Study Treatment Discontinuation visit
  - For subjects who attended the last on-treatment visit, use the Visit 8 (Week 24) date.
  - For subjects who died and did not attend a Study Treatment Discontinuation visit or the last on-treatment visit, use the date of death
  - For all other subjects, use the last recorded exposure start or stop date.
- If a subject's overall exposure start date is missing then it will be assumed to be their Day 1 visit date.
- If a subject received a treatment other than the randomised treatment during the study, the exposure will still be calculated based on overall exposure start and stop dates.

#### **Adverse Events**

- The most frequent on-treatment AEs will be defined as the on-treatment AEs experienced by 3
   % (after rounding) or more of subjects in any treatment group.
  - AE groups of special interest have been defined as AEs which have specified areas of
    interest for UMEC. The following table presents the special interest AE groups and
    subgroups. The complete list, including the PTs which contribute to each of the groups will
    be provided by Global Clinical Safety and Pharmacovigilance (GCSP) using the MedDRA
    version current at the time of reporting. This will be finalized prior to unblinding.

| Special Interest AE Group | Special Interest AE Subgroup |
|---|---|
| Cardiovascular effects | Cardiac Arrhythmia Cardiac Failure Cardiac Ischaemia Hypertension Stroke |
| Urinary Retention | |
| Pneumonia | |
| Anticholinergic syndrome | |
| Gastrointestinal obstruction | |
| Hypersensitivity | |
| LRTI excluding pneumonia | |
| Ocular effects (antimuscarinic) | |
| Paradoxical bronchospasm | |
| gallbladder disorders | |

- A flag will be derived to identify on-treatment AEs of special interest. In order to ensure
  consistency with the umeclidinium Global ISS, all outputs will use the same MedDRA version
  (i.e. v 15.0) and the same list of special interest terms as was used for the umeclidinium Global
  ISS.
- The AESI category designated as Pneumonia and LRTI will include lower respiratory tract infections and related diseases. Also, the category designated as "Anticholinergic Syndrome" will be referenced as "Anticholinergic Effects" since the Anticholinergic Syndrome SMQ which was used to located terms includes events that are often associated with anticholinergic or antimuscarinic medication, but are not necessarily diagnostic for anticholinergic syndrome.

#### **Laboratory Parameters**

• The baseline value for a parameter will be the most recent recorded value for that parameter before dosing on Day 1 at schedule visit.

#### **Laboratory Parameters**

- Laboratory data values will be classified as 'low', 'normal' or 'high' with reference to normal ranges.
- An 'any visit post-baseline' classification will be derived, in which subjects will be counted in the
  'low' and 'high' categories if they reported a low or high value at any scheduled, unscheduled or
  EW visit made after the start of study treatment, up to a maximum of two weeks after the last
  dose of study treatment. Subjects who did not report a low or high value at any visit after the
  start of study treatment will be counted in the 'normal' category.
- Change from baseline values will be classified relative to the normal range as 'to low', 'to
  normal or no change' or 'to high'. Subjects who do not change categories or move from out-ofrange to normal will be classified as 'to normal or no change'.
- An 'any visit post-baseline' change classification will be derived, in which subjects will be counted in the 'to low' and 'to high' categories if they reported a change from a 'normal' baseline to a value below or above the normal range (respectively) at any scheduled, unscheduled or EW visit made after the start of study treatment, up to a maximum of 2 weeks after the last dose of study treatment. Subjects who did not report a change to a value outside the normal range at any visit after the start of study treatment will be counted in the 'to normal or no change' category.
- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - $\circ$  Example 3: 0 Significant Digits = '< x' becomes x 1

#### **Vital Signs**

- The baseline value for a vital sign endpoint will be the most recent recorded value for that endpoint before dosing on Day 1 at schedule visit.
- The 'maximum/minimum post-baseline' value will be the maximum value for pulse rate and systolic blood pressure, or the minimum value for diastolic blood pressure, recorded at any scheduled, unscheduled or EW visit made after the start of study treatment.

#### 12-Lead ECG

- The baseline value for an ECG endpoint will be the most recent recorded value for that endpoint before dosing on Day 1 at schedule visit.
- A 'maximum post-baseline' QTc(F), QTc(B), PR interval and heart rate value will be derived as
  the maximum value recorded at any scheduled, unscheduled or EW visit made after the start of
  study treatment.
- QTc(F) values (including 'maximum post-baseline') will be categorised as follows:
  - ≤ 450 msec
  - $> 450 \text{ to} \le 480 \text{ msec}$
  - $> 480 \text{ to} \le 500 \text{ msec}$

#### 12-Lead ECG

- > 500 msec.
- Change from baseline QTc(F) values (including change to 'maximum post baseline') will be categorised as follows:
  - < -60 msec
  - ≥ -60 to < -30 msec
  - ≥ -30 to < 0 msec
  - ≥ 0 to < 30 msec
  - $\geq$  30 to < 60 msec
  - ≥60 msec.
- An 'any time post-baseline' ECG interpretation will be derived as the worst interpretation recorded at a scheduled, unscheduled or EW visit made after the start of study treatment.
   The order of severity from worst to best for ECG interpretation is: abnormal: clinically significant, abnormal: not clinically significant, normal, unable to interpret.
- Any ECG abnormality recorded by a subject with an ECG interpretation of 'abnormal: clinically significant' after the start of study treatment will be included in an 'any-time post-baseline' record of ECG abnormalities.
- Any ECG abnormality recorded by a subject after the start of study treatment will be included in an 'any-time post-baseline' record of all ECG abnormalities.

#### 10.6.4. Health- Related Quality of Life

#### St. George's Respiratory Questionnaire

- The SGRQ contains 76 items grouped into three domains (Symptoms, Activity and Impacts). The domain score will be calculated as the sum of the weighted scores for the non-missing items within each domain, dividing by the maximum possible score for those non-missing items and multiplying by 100. The SGRQ total score will be calculated as the sum of the weighted scores from all 76 items and dividing by the maximum possible score for the SGRQ and multiplying by 100. This calculation is outlined in the developer's guide (St. George's Respiratory Questionnaire Manual, 2009).
- If a subject has more than one response to a given item at a particular time point then the
  response will be taken as the average of the responses prior to calculating domain and total
  scores.
- If a subject has given both responses to a dichotomous question (yes/ no, true/false) the response to that question will be set to missing.
- If more than 25 % of items are missing from a domain, then the domain total will be set to
  missing. This equates to no more than two missed questions for the Symptom domain, no more
  than four missed questions for the Activity domain and no more than six missed questions for
  the Impacts domain. If any domain score is missing, then the total score will be set to missing.
- If the language of the SGRQ conducted during the study is different to the language used at Day 1, all SGRQ scores will be set to missing.
- The baseline SGRQ domain and total scores are those recorded on Day 1.
- A subject will be considered a 'responder' according to his SGRQ total score at each visit if the
  difference from the visit score to the baseline score was -4 units or lower. A subject will be

#### St. George's Respiratory Questionnaire

considered a 'non-responder' if the difference from the visit score to the baseline score was greater than -4 units.

 For the classification of responders, subjects with missing SGRQ total scores will be handled as detailed in Section 10.7.2.1 (Handling of Missing Responder).

#### CAT

- The CAT consists of eight items each formatted as a six-point differential scale: 0 (no impact) to 5 (high impact). A CAT score will be calculated by summing the non-missing scores on the eight items. If one or two items are missing, then the score for those items is set as the average of the non-missing items. If more than two items are missing, then the CAT score will be set to missing.
- The baseline CAT score will be that recorded on Day 1.
- A subject will be a responder if their on-treatment CAT score has decreased at least 2 units from baseline CAT total score.
- A subject will be considered a non-responder if their on-treatment CAT score has decreased by less than 2 units, has not changed, or has increased compared to baseline.
- For the classification of responders will be handled as detailed in Section 10.7.2.1 (Handling of Missing Responder).

#### **Healthcare Resource Utilisation**

 The total number of visits for each type of healthcare contact (telephone contacts, home visits (day), home visits (night), office/practice visits, urgent care/outpatient clinic visits, emergency room visits and the number of days in intensive care and in general hospital wards will be derived.

#### 10.6.5. Efficacy

#### Post-ipratropium FEV1

• The difference between post-ipratropium FEV1 and pre-salbutamol FEV1 will be calculated.

#### Reversibility and GOLD Stage

- A subject's responsiveness to salbutamol at Screening will be classified as 'Reversible' or 'Nonreversible' based on the difference between their pre-salbutamol assessment of FEV1 and their post-salbutamol assessment of FEV1 as follows:
  - o Reversible, if they had an difference in FEV1 of ≥12 % and ≥200 mL, or
  - Non-reversible, if they had a difference in FEV1 of < 200 mL or a ≥200 mL difference that was <12 % of the pre-salbutamol FEV1.</li>
- A subject's responsiveness to salbutamol and ipratropium at Screening will be classified as 'Reversible' or 'Non-reversible' based on the difference between their pre-salbutamol assessment of FEV1 and their post-ipratropium assessment of FEV1 as follows:
  - o Reversible, if they had a difference in FEV1 of ≥12 % and ≥200 mL, or
  - Non-reversible, if they had a difference in FEV1 of < 200 mL or a ≥200 mL difference that</li>

- was < 12 % of the pre-salbutamol FEV1.
- Subjects will be classified according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage (GOLD classification, [GOLD, 2011]): defined using the post-salbutamol percent predicted FEV1 assessed at Screening (Visit 1). Subjects will be classified as:
  - GOLD1: Mild FEV1 ≥80% predicted
  - GOLD 2: Moderate 50% ≤FEV1 < 80% predicted</li>
  - GOLD3: Severe 30% ≤FEV1 < 50% predicted</li>
  - GOLD4: Very Severe FEV1 <30% predicted</li>

#### **Trough FEV1 and FVC**

• The trough value for FEV1 and FVC at each of Days 2, 28, 56, 84, 112, 168 and 169 is calculated from the values at the assessments made 23 h and 24 h after dosing on the previous day. If the actual time of an assessment is after the time of dosing on the current day, the value will not be used in the calculation of trough. For the PP population, a value will additionally be excluded from the trough calculation if the assessment is outside the time window of 22.5-24.5 h after dosing on the previous day (see Section 10.1.2 (Exclusions of Data from Per Protocol Analyses)). If one of the values is missing or excluded then the trough will be the single remaining value; otherwise the trough will be the mean of the two values.

#### BDI/TDI

- The baseline dyspnoea index (BDI) focal score will be calculated as the sum of the ratings recorded for each of the three individual scales (Baseline Functional Impairment, Baseline Magnitude of Task, Baseline Magnitude of Effort). Each of these scales has five possible scores ranging from 0 to 4 (with lower scores indicating more impairment), so the range of the BDI focal score is 0 to 12. If a score is missing (or has a value of W, X or Y) for any of the three scales, then the BDI focal score will be set to missing.
- The TDI focal score will be calculated as the sum of the ratings recorded for each of the three individual scales (Change in Functional Impairment, Change in Magnitude of Task, Change in Magnitude of Effort). Each of these scales has seven possible scores ranging from -3 (major deterioration) to +3 (major improvement), so the range of the TDI focal score is -9 to +9. If a score is missing (or has a value of Z) for any of the three scales, then the TDI focal score will be set to missing.
- A subject will be considered a 'responder' according to TDI at each visit if the TDI focal score
  was at least 1 unit at that visit. A subject will be considered a 'non-responder' if the score was
  less than 1 unit.
- For the classification of responders, subjects with missing TDI assessments will be handled as detailed in Section 10.7.2.1 (Handing of Missing Responder).

#### Weighted Mean FEV1 and FVC

- Weighted mean FEV1 and FVC will be calculated over the nominal 0-6 h post dose period.
   Values from post-dose assessments which are actually before the time of dosing will be excluded from the calculation.
- The 0 h value is the average value obtained 30 min and 5 min pre-dose, and both the 0 h and 6 h values must be present for a 0-6 h weighted mean to be calculated.
- The 0-6 h weighted mean will be derived by calculating the area under the FEV1 or FVC/time

#### Weighted Mean FEV1 and FVC

curve over the nominal time points of 0 h (as defined above), 15 and 30 min, 1, 3 and 6 h, using the trapezoidal rule, and then dividing by the actual time between dosing and the 6 h assessment. For post-dose observations the actual time of assessment relative to the time of dosing will be used for the calculation.

Weighted Mean (0-6h) = 
$$\left[\frac{1}{2}\sum_{i=1}^{I-1}(t_{i+1}-t_i)(y_i+y_{i+1})\right]/[t_I-t_f]$$

#### where

y<sub>i</sub> represents the value of the endpoint at the ith timepoint,

t<sub>i</sub> represents the actual relative time at the ith timepoint,

 $t_f$  represents the actual relative time at the first timepoint ( $t_f$  = 0 as the pre-dose measurement is used),

t<sub>1</sub> represents the actual relative time at the last timepoint (the 6h timepoint),

I represents the number of timepoints used in the AUC calculation.

If missing values are present in data required for the calculation of the weighted means, the following approach will be employed:

- If more than a third of the observations are missing then the weighted mean will be set to missing for that subject.
- If an observation is missing between two non-missing observations, the value will be interpolated between the two non-missing values.
- If there are two or more missing points that occur consecutively then the weighted mean will be set to missing.
- If the first time-point is missing then the weighted mean will be set to missing.
- If the last time-point is missing then the weighted mean will be set to missing.

#### **Rescue Use**

- For rescue use, 'day' refers to the period (24 hours) between one record of rescue use and the next in the database.
- The total puffs of rescue for each day will be calculated as number of salbutamol puffs. If the number of puffs are missing then the total puffs will be set to missing for that day.
- Rescue use will be summarised over the periods defined in below table:

| Period | First day | Last day |
|---|---|---|
| Baseline | Latest of 6 days before Visit 2 and day after Visit 1 | Day of Visit 2 |
| Week 1-4 | Study day 2 (day after Visit 2) | Study day 29 |
| Week 5-8 | Study day 30 | Study day 57 |

| Res | cue Use | | |
|---|---|---|---|
| | Week 9-12 | Study day 58 | Study day 85 |
| | Week 13-16 | Study day 86 | Study day 113 |
| | Week 17-20 | Study day 114 | Study day 141 |
| | Week 21-24 | Study day 142 | Earliest of Study day 169 and day before Visit 9 |
| | Week 1-24 | Study day 2 (day after Visit 2) | Earliest of Study day 169 and day before Visit 9 |

- For each summary period, the mean number of puffs per day and the percentage of rescue-free days will be calculated, provided at least half the days within the summary period have nonmissing values for the endpoint.
- Any data recorded after study day 169 (but before Visit 9) will not be included in any summaries.

#### Time to Onset on Day 1

- The time to onset on Day 1 is calculated as the time (both nominal and actual) that the first post-dose FEV1 during the 0-6 h post-dose period is ≥100 mL above baseline FEV1. Post-dose assessments that are actually pre-dose will be considered missing in the calculation.
- Subjects who have at least one FEV1 assessment within the 0-6 h post-dose period but do not achieve a ≥100 mL increase from baseline over 0-6 h post-dose will be considered censored.

# Increase in FEV1 of ≥12% and ≥200 mL above Baseline at any Time During 0-6 h Post-dose on Day 1

- A flag will be derived to identify whether or not a subject achieved an increase in FEV1 of ≥12% and ≥200 mL above baseline at any time during 0-6 h post-dose on Day 1. The flag will have values as follows:
  - 1, if any FEV1 value recorded at 15 or 30 min, 1, 3 or 6 h was ≥12 % and ≥200 mL above baseline.
  - 0, if no FEV1 value recorded at 15 or 30 min, 1, 3 or 6 h was ≥12 % and ≥200 mL above baseline.

#### Increase of ≥100 mL above Baseline in Trough FEV1

- A flag will be derived to identify whether or not a subject achieved an increase of ≥100 mL above baseline in trough FEV1 at each of Days 2, 28, 56, 84, 112, 168 and 169. The flag will have values as follows:
  - o 1, if the trough FEV1 was ≥100 mL above baseline.
  - 0, if the trough FEV1 was < 100 mL above baseline, or the trough FEV1 was missing with no subsequent non-missing trough FEV1 values.
  - Missing, if the trough FEV1 was missing but subsequent trough FEV1 values were nonmissing.

# 10.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

## 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as on completion of final on-treatment clinic visit (Visit 9).</li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |
| | <ul> <li>In general, the minimum data required will be a baseline evaluation and at least one post-baseline evaluation.</li> <li>If a subject withdraws at a scheduled treatment visit, then any data collected at that visit associated with scheduled visit procedures will be used (under the scheduled visit assignment) in all summaries and analyses wherever possible.</li> <li>All other data collected as part of the early withdrawal at a scheduled visit, or at a standalone EW visit, will only be used in summary or analysis tables as part of the 'worst case post baseline' summary/analysis.</li> </ul> |
| | Early withdrawal data will be included in any relevant listing. |

# 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | For efficacy endpoints, missing data is expected to arise mainly from subjects missing complete visits or time points. |
| | <ul> <li>The amount of occasional missing data for covariates included in the statistical<br/>analysis is expected to be minimal. Missing data will not be directly imputed in<br/>primary analysis of each endpoint.</li> </ul> |
| | <ul> <li>For analysis of trough FEV1 at Day 169, sensitivity analyses with LOCF will be<br/>produced for supportive analysis.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.7.2.1. Handling of Missing Responder

| Element | Reporting Detail |
|---|---|
| Responder | <ul> <li>Subjects with missing data and a subsequent non-missing assessment will not be considered a responder or non-responder but will be left as missing.</li> <li>Subjects with missing data and no subsequent assessments will be considered a non-responder.</li> </ul> |
| | No extra visits will be added and no imputation performed in the original dataset. |
| | The analysis dataset will initially contain rows for each visit at which at least one |

| Element | Reporting Detail |
|---|---|
| | derived variable (excluding baseline) is able to be calculated. For these rows, IMPFLAG will be 1 (not imputed). |
| | <ul> <li>For subjects who do not provide data at the final visit, additional rows will be<br/>created for each subsequent visit after their final visit (i.e. their time of<br/>withdrawal) with non-missing data which is planned to be included in the<br/>responder analysis. For these rows, IMPFLAG will be 0 (imputed) and<br/>responder status will be 'Non-responder'.</li> </ul> |
| | <ul> <li>If the final visit containing non-missing data does not provide enough data to calculate the derived variable on which the responder status is based (e.g. some domains of the SGRQ are present but not all, so the total score cannot be created), then IMPFLAG will be changed to 0 (imputed) and responder status will be 'Non-responder' on that row.</li> </ul> |
| | <ul> <li>Apart from derived FEV1 and FVC, the listings should not contain any rows where all the derived variables are missing, except for the rows which are imputed. (The FEV1 listing may have a blank row between two non-missing rows because all FEV1 derived variables are missing but FVC derived variables are present – IMPFLAG should still be 1 for these rows.)</li> </ul> |
| | <ul> <li>If the baseline value is missing, or there are no post-baseline non-missing<br/>assessments, no imputation will be performed</li> </ul> |
| | <ul> <li>No visits will be imputed if they are between two visits with non-missing assessments</li> </ul> |

# 10.7.2.2. Handing of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |

# 10.7.2.3. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> </ul> </li> </ul> |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 10.7.2.4. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| MMRM | Missing data will not be directly imputed in this analysis; however, all non-missing data for a subject will be used within the analysis to estimate the treatment effect |
| ANCOVA | <ul> <li>For analysis of trough FEV1 at Day 169, sensitivity analyses with LOCF to imputed missing data will be produced for supportive analysis.</li> <li>Missing data will not be imputed for other analysis.</li> </ul> |
| Cox's proportional Analysis | Missing data will not be imputed. |
| Logistic regression Analysis | Missing data will not be imputed. |

# 10.8. Appendix 8: Values of Potential Clinical Importance

## 10.8.1. Laboratory Values

Threshold values for liver function test results, which are considered values of potential clinical importance, are:

- 3 times the upper limit of normal (ULN) for Alanine Aminotransferase (ALT)
- 2 times the ULN for Total Bilirubin (BILT).

Graphical displays of liver function test results will be produced as described in Section 8.2 (Clinical Laboratory Analyses) to identify any results above the thresholds.

Laboratory values will be flagged relative to the normal range. Clinical concern ranges will not be used.

#### 10.8.2. ECG

Clinical concern ranges will not be used.

#### 10.8.3. Vital Signs

Clinical concern ranges will not be used.

# 10.9. Appendix 9: Multicenter Studies

This study was randomized centrally within country. No strata were defined.

Country will be considered a fixed effect in all analyses on overall population. For primary efficacy analysis, interaction with treatment will be explored by fitting a model with an additional treatment by country interaction term; any interaction found to be statistically significant at the 10 % level will be further investigated and characterised. Center will not be included as a covariate in China subgroup statistical analyses.

All results will be produced for all countries combined. In addition, summary statistics of demography, screening lung function, primary and secondary endpoints will be produced by country.

# 10.10. Appendix 10: Examination of Covariates, Subgroups & Other Strata

The details of covariates that will be used in statistical analyses have been clarified in Section 7.1 (Primary Statistical Analyses), Section 7.2 (Secondary Statistical Analyses) and Section 7.3 (Other Statistical Analyses).

Consistency of treatment effect across covariates fitted in the primary efficacy endpoint analysis models will be examined by fitting separate models to examine treatment by baseline, treatment by country (not done for China alone sub-group analysis) and treatment by smoking status at screening interactions. Separate analysis models will also be fitted to examine treatment by ICS use, treatment by reversibility to salbutamol and treatment by percent predicted  $FEV_1$ .

No formal statistical analysis of sub-groups of the study population for either the overall analysis or the China subgroup analysis will be performed.

# 10.11. Appendix 11: Multiple Comparisons & Multiplicity

There is no adjustment for multiplicity to be applied in this study for the analysis on all countries overall as there is only one primary endpoint (Clinic visit trough (prebronchodilator) FEV1 on Treatment Day 169) and only one primary comparison (UMEC62.5 mcg vs. placebo) of interest. Treatment comparisons for secondary and other endpoints will be considered exploratory.

For China subgroup analysis, as the China subgroup analysis is powered, the inference on the primary endpoint on China subgroup is dependent on statistical significance having been achieved for the primary endpoint on the analysis on all countries overall. Treatment comparisons for secondary and other endpoints in China subgroup analysis will also be considered exploratory.

# 10.12. Appendix 12: Model Checking and Diagnostics for Statistical Analyses

#### 10.12.1. Statistical Analysis Assumptions

| Endpoint(s) | Trough FEV1 |
|-------------|-----------------|
| | Trough FVC |
| | TDI Focal Score |
| | Serial FEV1 |
| | Serial FVC |
| Analysis | MMRM |

- O The Kenward and Roger method (KR) for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
  - O In the event the model fails to run using the KR method, then the residual method will be used instead.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

# Endpoint(s) O-6 h weighted mean FEV1 on Day 1 Mean number of puffs of rescue medication per day over each treatment period Pulse rate Systolic Diastolic blood pressure QTc(F) PR interval Heart rate Analysis ANCOVA

Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

| Endpoint(s) | <ul> <li>Time to Onset (an increase of 100mL in FEV1 above baseline) during 0-6 h post-dose on Day 1</li> <li>Time to First COPD Exacerbation</li> </ul> |
|---|---|
| Analysis | Cox's proportional hazards model |
| The n | proportional hazards assumption for this method of analysis will be examined by |

The proportional hazards assumption for this method of analysis will be examined by obtaining the Kaplan-Meier estimates of the survival function S(t) over time separately for treatment group. Under the assumption of proportional hazard between the treatment

groups, In{-In[S(t)]} for the two groups should be parallel to each other and the distance between them constant. If the curves are approximately parallel, then the proportional hazard assumption is not violated. If these curves cross each other or diverge greatly from the assumption of parallel lines, then the assumption is not met.

| Endpoint(s) | • Proportion Achieving Increase in FEV1 of ≥12 % and ≥200 mL above Baseline at any Time During 0-6 h Post-dose on Day 1 |
|---|---|
| | • Proportion Achieving Increase of ≥ 100 mL above Baseline in Trough FEV1 |
| | <ul> <li>Proportion of Responders According to TDI Focal Score</li> </ul> |
| Analysis | Logistic regression model |

- Computation of confidence intervals for the odds ratios is based on the individual Wald tests.
- BUD/FOR will be used as the reference level for treatment
- Goodness-of-fit of the logistic model will be examined using the LACKFIT option for the model statement in SAS. Index plots of the Pearson residuals and deviance criteria residuals will be plotted by using the IPLOTS option for the model statement in SAS.

# 10.13. Appendix 13 – Abbreviations & Trade Marks

# 10.13.1. Abbreviations

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| GUI | Guidance |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| GSK | GlaxoSmithKline |

# 10.13.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| HARP |
| RAMOS |
| RANDALL |

| Trademarks not<br>owned by the<br>GlaxoSmithKline<br>Group of Companies |
|-------------------------------------------------------------------------|
| SAS |
| S-PLUS |

# 10.14. Appendix 14: List of Data Displays

## 10.14.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|--------------------------------------------|-------------|-------------|
| Study Population (Overall Analysis) | 1.1 to 1.37 | 1.1 to 1.1 |
| Study Population (China Subgroup Analysis) | 1.1 to 1.35 | 1.1 to 1.1 |
| Efficacy(Overall Analysis) | 2.1 to 2.56 | 2.1 to 2.21 |
| Efficacy (China Subgroup Analysis) | 2.1 to 2.49 | 2.1 to 2.21 |
| Safety (Overall Analysis) | 3.1 to 3.48 | 3.1 to 3.17 |
| Safety (China Subgroup Analysis) | 3.1 to 3.48 | 3.1 to 3.17 |
| Section | List | ings |
| ICH Listings | 1 to | 25 |
| Other Listings | 26 t | o 54 |

# 10.14.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 15: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|----------|--------|-------|---------|
| Efficacy | NA | NA | EFF_L1 |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 10.14.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC [1] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 10.14.4. Study Population Tables

| Study I | Study Population Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 1.1. | 1.1. | All Subjects<br>Enrolled | DB2114634<br>5.01 | Summary of Subject Populations | | SAC |
| 1.2. | 1.2. | Modified ITT | DB2114634<br>5.09 | Summary of Exclusions from the Per Protocol Analysis | | SAC |
| 1.3. | 1.3. | Modified ITT | DB2114634<br>5.02 | Summary of Attendance at Each Clinic Visit | | SAC |
| 1.4. | 1.4. | Modified ITT | DB2114634<br>5.03 | Summary of Subject Disposition | | SAC[1] |
| 1.5. | 1.5. | Screen and<br>Run-in Failure | DB2114634<br>5.04 | Summary of Reasons for Screen Failures | | SAC |
| 1.6. | 1.6. | Screen and<br>Run-in Failure | DB2114634<br>5.05 | Summary of Reasons for Run-in Failures | | SAC |
| 1.7. | 1.7. | Modified ITT | DB2114634<br>5.06 | Summary of Number of Subjects by Country and Centre | For China subgroup,<br>Country will be omitted<br>from the title. | SAC |
| 1.8. | 1.8. | Screen and<br>Run-in Failure | DB2114634<br>5.07 | Summary of Inclusion/Exclusion/Randomisation Criteria Deviations for Screen or Run-in Failures | | SAC |
| 1.9. | 1.9. | Modified ITT | DB2114634<br>5.08 | Summary of Inclusion/Exclusion/Randomisation Criteria Deviations for Modified Intent-to-treat Subjects | | SAC |

| Study Population Tables | | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 1.10. | 1.10. | Modified ITT | DB2114634<br>5.09 | Summary of Important Protocol Deviations | Remove rows of Full Protocol Deviations, Partial Protocol Deviations and Timepoint Specific Protocol Deviations and summarize all PDs with DVIMPFL marked as "Y". | SAC |
| 1.11. | 1.11. | Modified ITT | DB2114634<br>5.10 | Summary of Demographic Characteristics | | SAC[1] |
| 1.12. | NA | Modified ITT | DB2114634<br>5.11 | Summary of Demographic Characteristics by Country | | SAC |
| 1.13. | 1.12. | PP | DB2114634<br>5.12 | Summary of Demographic Characteristics | | SAC |
| 1.14. | 1.13. | Modified ITT | DB2114634<br>5.13 | Summary of Race and Racial Combinations | | SAC |
| 1.15. | 1.14. | Modified ITT | DB2114634<br>5.14 | Summary of Race and Racial Combination Details | | SAC |
| 1.16. | 1.15. | Modified ITT | DB2114634<br>5.15 | Summary of Current Medical Conditions | | SAC |

| Study Population Tables | | | | | | | | | | |
|---|---|---|---|---|---|---|--|--|--|--|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] | | | | |
| 1.17. | 1.16. | Modified ITT | DB2114634<br>5.16 | Summary of Past Medical Conditions | | SAC | | | | |
| 1.18. | 1.17. | Modified ITT | DB2114634<br>5.17 | Summary of Past Cholecystectomies | | SAC | | | | |
| 1.19. | 1.18. | Modified ITT | DB2114634<br>5.18 | Summary of Family History of Cardiovascular Risk Factors | | SAC | | | | |
| 1.20. | 1.19. | Modified ITT | DB2114634<br>5.19 | Summary of COPD History | | SAC | | | | |
| 1.21. | 1.20. | Modified ITT | DB2114634<br>5.20 | Summary of COPD Exacerbation History | | SAC | | | | |
| 1.22. | 1.21. | Modified ITT | DB2114634<br>5.21 | Summary of Smoking History | | SAC | | | | |
| 1.23. | 1.22. | Modified ITT | DB2114634<br>5.22 | Summary of Smoking Status | | SAC | | | | |
| 1.24. | 1.23. | Modified ITT | DB2114634<br>5.23 | Summary of Screening Lung Function Test Results | | SAC | | | | |
| 1.25. | NA | Modified ITT | DB2114634<br>5.24 | Summary of Screening Lung Function Test Results by Country/Region | | SAC | | | | |
| Study I | Study Population Tables | | | | | | | | |
|---|---|---|---|---|---|---|--|--|--|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] | | | |
| 1.26. | 1.24. | Modified ITT | DB2114634<br>5.25 | Summary of GOLD Stage, Percentage of Reversible Subjects and ICS Use at Screening | | SAC | | | |
| 1.27. | 1.25. | Modified ITT | DB2114634<br>5.26 | Summary of mMRC Dyspnoea Scale | | SAC | | | |
| 1.28. | 1.26. | Modified ITT | DB2114634<br>5.27 | Summary of COPD Concomitant Medications Not Given for an Exacerbation Taken Pre-treatment | | SAC | | | |
| 1.29. | 1.27. | Modified ITT | DB2114634<br>5.28 | Summary of COPD Concomitant Medications Not Given for an Exacerbation Taken On-treatment | | SAC | | | |
| 1.30. | 1.28. | Modified ITT | DB2114634<br>5.29 | Summary of COPD Concomitant Medications Not Given for an Exacerbation Taken Post-treatment | | SAC | | | |
| 1.31. | 1.29. | Modified ITT | DB2114634<br>5.30 | Summary of Concomitant Medications Given for an<br>Exacerbation Taken Pre-treatment | | SAC | | | |
| 1.32. | 1.30. | Modified ITT | DB2114634<br>5.31 | Summary of Concomitant Medications Given for an<br>Exacerbation Taken On-treatment | | SAC | | | |
| 1.33. | 1.31. | Modified ITT | DB2114634<br>5.32 | Summary of Concomitant Medications Given for an<br>Exacerbation Taken Post-treatment | | SAC | | | |
| 1.34. | 1.32. | Modified ITT | DB2114634<br>5.33 | Summary of Non-COPD Concomitant Medications Taken Pre-treatment | | SAC | | | |

| Study I | Study Population Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 1.35. | 1.33. | Modified ITT | DB2114634<br>5.34 | Summary of Non-COPD Concomitant Medications Taken<br>On-treatment | | SAC |
| 1.36. | 1.34. | Modified ITT | DB2114634<br>5.35 | Summary of Non-COPD Concomitant Medications Taken Post-treatment | | SAC |
| 1.37. | 1.35. | Modified ITT | DB2114634<br>5.36 | Summary of Overall Percentage Treatment Compliance | | SAC |

# 10.14.5. Study Population Figures

| Study P | Study Population: Figures | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | SUDOMOUD PANILISTIAN | | | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.1 | 1.1 | Modified ITT | DB2114634<br>5.01 | Subject Withdrawals over Time | | SAC |

### 10.14.6. Efficacy Tables

| Efficacy: | Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | Example Shell Output | | Programming<br>Notes | Deliverable<br>[Priority] |
| 21 21 Modified ITT | | DB2114634<br>6.01 | Summary of Baseline FEV1 (L), Modified Intent-to-treat | | SAC[1] | |
| 2.2. | NA | Modified ITT | DB2114634<br>6.02 | Summary of Baseline FEV1 (L) by Country/Region, Intent-to-treat | | SAC |
| 2.3. | 2.2 | Modified ITT DB2114634 Summary of Trough FEV1 (L), Modified Intent-to-treat 6.03 | | SAC[1] | | |
| 2.4. | NA | Modified ITT | DB2114634<br>6.04 | Summary of Trough FEV1 (L) by Country/Region, Modified Intent-to-treat | | SAC |
| 2.5. | 2.3 | Modified ITT | DB2114634<br>6.05 | Analysis of Trough FEV1 (L), Modified Intent-to-treat, Repeated Measures | | SAC[1] |
| 2.6. | 2.4 | PP | DB2114634<br>6.06 | Summary of Baseline FEV1 (L), Per Protocol | | SAC |
| 2.7. | NA | PP | DB2114634<br>6.07 | Summary of Baseline FEV1 (L) by Country/Region, Per Protocol | | SAC |
| 2.8. | 2.5 | PP | DB2114634<br>6.08 | Summary of Trough FEV1 (L), Per Protocol | | SAC |
| 2.9. | NA | PP DB2114634 Summary of Trough FE Protocol | | Summary of Trough FEV1 (L) by Country/Region, Per Protocol | | SAC |
| 2.10. | 2.6 | | | | SAC | |

| Efficacy: | : Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | Example Shell IITIE No | | Programming<br>Notes | Deliverable<br>[Priority] |
| 2.11. | 2.11. 2.7 Modified I | | HZC113684<br>6.07 | Summary of Trough FEV1 (L) at Day 169 LOCF | | SAC |
| 2.12. | 2.8 | Modified ITT | HZC113684<br>6.08 | Statistical Analysis of Trough FEV1 (L) at Day 169 using LOCF | | SAC |
| 2.13. | 2.9 | Modified ITT | DB2114634<br>6.11 | Summary of 0-6 h Weighted Mean FEV1 (L) | | SAC |
| 2.14. | NA | Modified ITT | DB2114634<br>6.12 | Summary of 0-6 h Weighted Mean (L) by Country/Region | | SAC |
| 2.15. | 2.10 | Modified ITT | DB2114634<br>6.13 | Analysis of 0-6 h Weighted Mean FEV1 (L) | | SAC |
| 2.16. | 2.11 | Modified ITT | DB2114634<br>6.14 | Summary of Time to Onset (an increase of 100mL in FEV1 above baseline) on Day 1 | | SAC |
| 2.17. | 2.12 | Modified ITT | DB2114634<br>6.15 | Analysis of Time to Onset (min) (an increase of 100mL in FEV1 above baseline) on Day 1 | | SAC |
| 2.18. | 2.13 | Modified ITT DB2114634 6.16 | | Summary and Analysis of Proportion of Subjects Achieving Increase in FEV1 of >= 12 % and >= 200 mL above Baseline at Any Time during 0-6 h Post-dose on Day 1 | | SAC |
| 2.19. | 2.14 | Modified ITT | DB2114634<br>6.17 | Summary and Analysis of Proportion of Subjects Achieving Increase in Trough FEV1 of >= 100 mL above Baseline | | SAC |
| 2.20. | 2.15 | Modified ITT | DB2114634<br>6.18 | Summary of Serial FEV1 (L) | | SAC |

| Efficacy | Efficacy: Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | Example Shell No. | | Programming<br>Notes | Deliverable<br>[Priority] |
| 2.21. | 2.16 | Modified ITT | DB2114634<br>6.19 | Summary of Change from Baseline in Serial FEV1 (L) | | SAC |
| 2.22. | 2.17 | Modified ITT | DB2114634<br>6.20 | Analysis of Serial FEV1 (L) on Day 1 | | SAC |
| 2.23. | 2.18 | Modified ITT | DB2114634<br>6.21 | Summary of Baseline FVC (L) | | SAC |
| 2.24. | 2.19 | 2.19 Modified ITT DB2114634 Summary of Trough FVC (L) 6.22 | | | SAC | |
| 2.25. | 2.20 | 20 Modified ITT DB2114634 Analysis of Trough FVC (L) 6.23 | | | SAC | |
| 2.26. | 2.21 | Modified ITT | DB2114634<br>6.24 | Summary of Serial FVC (L) | | SAC |
| 2.27. | 2.22 | Modified ITT | DB2114634<br>6.25 | Summary of Change from Baseline in Serial FVC (L) | | SAC |
| 2.28. | 2.23 | Modified ITT | DB2114634<br>6.26 | Analysis of Serial FVC (L) on Day 1 | | SAC |
| 2.29. | 2.24 | Modified ITT | DB2114634<br>6.27 | Summary of Percentage of Rescue-Free Days | | SAC |
| 2.30. | 2.25 | | | | SAC | |
| 2.31. | 2.26 | | | SAC | | |

| Efficacy | Efficacy: Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID /<br>Example Shell | Example Shell IIIIe | | Deliverable<br>[Priority] |
| 2.32. | 2.27 | Modified ITT | DB2114634<br>6.30 | Summary of BDI Focal Score | | SAC[1] |
| 2.33. | NA | Modified ITT | DB2114634<br>6.31 | Summary of BDI Focal Score by Country/Region | | SAC |
| 2.34. | 2.28 | Modified ITT | DB2114634<br>6.32 | Summary of TDI Focal Score | | SAC[1] |
| 2.35. | NA | Modified ITT | DB2114634<br>6.33 | Summary of TDI Focal Score by Country/Region | cal Score by Country/Region | |
| 2.36. | 2.29 | Modified ITT | DB2114634<br>6.34 | Analysis of TDI Focal Score, Repeated Measures | Repeated Measures | |
| 2.37. | 2.30 | Modified ITT | DB2114634<br>6.35 | Summary and Analysis of Proportion of Responders According to TDI | | SAC |
| 2.38. | 2.31 | Modified ITT | DB2114634<br>6.36 | Summary of Baseline SGRQ Scores | | SAC |
| 2.39. | 2.32 | Modified ITT | DB2114634<br>6.37 | Summary of SGRQ Total Score | | SAC |
| 2.40. | 2.33 | Modified ITT | DB2114634<br>6.38 | Summary of SGRQ Symptoms Domain Score | | SAC |
| 2.41. | 2.34 | Modified ITT | DB2114634<br>6.39 | Summary of SGRQ Activity Domain Score | | SAC |
| 2.42. | 2.35 | Modified ITT | DB2114634<br>6.40 | Summary of SGRQ Impacts Domain Score | | SAC |

| Efficacy | : Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | Example Shell | | Programming<br>Notes | Deliverable<br>[Priority] |
| 2.43. | 2.43. 2.36 Modified ITT | | DB2114634<br>6.41 | | | SAC |
| 2.44. | 2.37 | Modified ITT | DB2114634<br>6.42 | Summary and Analysis of Proportion of Responders<br>According to SGRQ Total Score | | SAC |
| 2.45. | 2.38 | Modified ITT DB2114634 Summary of Healthcare Resource Utilisation 6.43 | | SAC | | |
| 2.46. | 2.39 | Modified ITT | DB2114634<br>6.44 | 4 Summary of Baseline CAT Score | | SAC |
| 2.47. | 2.40 | Modified ITT | DB2114634<br>6.45 | Summary of CAT Score | | SAC |
| 2.48. | 2.41 | Modified ITT | DB2114634<br>6.41 | Analysis of CAT Score | | SAC |
| 2.49. | 2.42 | Modified ITT | DB2114634<br>6.42 | Summary and Analysis of Proportion of Responders<br>According to CAT Score up to Week 24 | | SAC |
| 2.50. | 2.43 | Modified ITT | DB2114634<br>6.46 | Summary of On-treatment COPD Exacerbations | | SAC |
| 2.51. | 2.44 | Modified ITT | DB2114634<br>6.47 | Summary of Post-treatment COPD Exacerbations | | SAC |
| 2.52. | 2.45 | Modified ITT | DB2114634 Summary and Analysis of Time to First On-treatment Exacerbation (days) | | SAC | |
| Stats Ap | pendix | | • | | | |
| 2.53. | 2.46 | Modified ITT | DB2114634<br>10.01 | Type III Tests of Fixed Effects for Repeated Measures Analysis of Trough FEV1 | | SAC |

| Efficacy | Efficacy: Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 2.54. | 2.47 | Modified ITT | DB2114634<br>10.02 | Covariance Parameter Estimates for Repeated Measures Analysis of Trough FEV1 | | SAC |
| 2.55. | 2.48 | Modified ITT | DB2114634<br>10.03 | Significance Levels for Interactions of Treatment with Smoking Status, country and Baseline for Trough FEV1 | | SAC |
| 2.56. | 2.49 | Modified ITT | DB2114634<br>10.04 | Significance Levels for Interactions of Treatment with ICS Use, Reversibility, Percent Predicted FEV1 for Trough FEV1 | | SAC |

## 10.14.7. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.1. | 2.1 | Modified<br>ITT | DB2114634<br>6.01 | Box Plot of Change from Baseline in Trough FEV1 (L) at Day 169 | | SAC |
| 2.2. | 2.2 | Modified<br>ITT | DB2114634<br>6.02 | Empirical Distribution Function Plot of Change from Baseline in Trough FEV1 (L) at Day 169 | | SAC |
| 2.3. | 2.3 | Modified<br>ITT | DB2114634<br>6.03 | Least Squares Mean (95% CI) Change from Baseline in Trough FEV1 (L), Modified Intent-to-treat | | SAC |
| 2.4. | 2.4 | Modified<br>ITT | DB2114634<br>6.04 | Least Squares Mean (95% CI) Treatment Differences from Placebo in Change from Baseline in Trough FEV1 (L), Modified Intent-to-treat | | SAC |
| 2.5. | 2.5 | PP | DB2114634<br>6.05 | Least Squares Mean (95% CI) Change from Baseline in Trough FEV1 (L), Per Protocol | | SAC |
| 2.6. | 2.6 | PP | DB2114634<br>6.06 | Least Squares Mean (95% CI) Treatment Differences from Placebo in Change from Baseline in Trough FEV1 (L), Per Protocol | | SAC |
| 2.7. | 2.7 | Modified<br>ITT | DB2114634<br>6.07 | Kaplan-Meier Estimates of Time to Onset (min) on Day 1 | | SAC |
| 2.8. | 2.8 | Modified<br>ITT | DB2114634<br>6.08 | Least Squares Mean (95% CI) Change from Baseline in FEV1 (L) Over Time on Day 1 | | SAC |
| 2.9. | 2.9 | Modified<br>ITT | DB2114634<br>6.09 | Least Squares Mean (95% CI) Treatment Differences from Placebo in Change from Baseline in FEV1 (L) Over Time on Day 1 | | SAC |
| 2.10. | 2.10 | Modified<br>ITT | DB2114634<br>6.10 | Least Squares Mean (95% CI) Change from Baseline in Trough FVC (L) | | SAC |

| Efficacy | Efficacy: Figures | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11. | 2.11 | Modified<br>ITT | DB2114634<br>6.11 | Least Squares Mean (95% CI) Treatment Differences from Placebo in Change from Baseline in Trough FVC (L) | | SAC |
| 2.12. | 2.12 | Modified<br>ITT | DB2114634<br>6.12 | Least Squares Mean (95% CI) Change from Baseline in FVC (L) Over Time on Day 1 | | SAC |
| 2.13. | 2.13 | Modified<br>ITT | DB2114634<br>6.13 | Least Squares Mean (95% CI) Treatment Differences from Placebo in Change from Baseline in FVC (L) Over Time on Day 1 | | SAC |
| 2.14. | 2.14 | Modified<br>ITT | DB2114634<br>6.14 | Least Squares Mean (95% CI) TDI Focal Score | | SAC |
| 2.15. | 2.15 | Modified<br>ITT | DB2114634<br>6.15 | Least Squares Mean (95% CI) Treatment Differences from Placebo in TDI Focal Score | | SAC |
| 2.16. | 2.16 | Modified<br>ITT | DB2114634<br>6.16 | Empirical Distribution Function of Change from Baseline in SGRQ Total Score at Day 168 | | SAC |
| 2.17. | 2.17 | Modified<br>ITT | DB2114634<br>6.17 | Least Squares Means (95% CI) Change from Baseline in SGRQ Total Score | | SAC |
| 2.18. | 2.18 | Modified<br>ITT | DB2114634<br>6.18 | Least Squares Mean (95% CI) Treatment Differences from Placebo in Change from Baseline in SGRQ Total Score | | SAC |
| 2.19. | 2.19 | Modified<br>ITT | DB2114634<br>6.19 | Time to First On-treatment COPD Exacerbation (days) | | SAC |
| 2.20. | 2.20 | Modified<br>ITT | DB2114634<br>6.20 | Scatter plot of Change from Baseline CAT scores versus<br>Change from Baseline Trough FEV1 at Day 168 | | SAC |

| Efficacy | Efficacy: Figures | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.21. | 2.21 | Modified<br>ITT | DB2114634<br>6.21 | Scatter Plot of Baseline CAT scores versus Baseline FEV1 | | SAC |

### 10.14.8. Safety Tables

| Safety : | Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.1. | 3.1 | Modified<br>ITT | DB2114634 | Summary of Exposure | | SAC |
| 3.2. | 3.2 | Modified<br>ITT | DB2114634<br>7.02 | Overview of Adverse Events | | SAC[1] |
| 3.3. | 3.3 | Modified<br>ITT | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.4. | 3.4 | Modified<br>ITT | AE3 | Summary of Common Adverse Events by Overall Frequency | A common AE is one reported by 3% or more of subjects in any treatment group | SAC |
| 3.5. | 3.5 | Modified<br>ITT | DB2114634<br>7.03 | Summary of On-treatment Adverse Events | | SAC |
| 3.6. | 3.6 | Modified<br>ITT | DB2114634<br>7.04 | Summary of Post-treatment Adverse Events | | SAC |
| 3.7. | 3.7 | Modified<br>ITT | DB2114634<br>7.05 | Summary of On-treatment Adverse Events Reported by 3 % (after rounding) or More Subjects in Any Treatment Group | | SAC |
| 3.8. | 3.8 | Modified<br>ITT | DB2114634<br>7.06 | Summary of On-treatment Common Non-serious Adverse Events | A common AE is one reported by 3% or more of subjects in any treatment group. | SAC |
| 3.9. | 3.9 | Modified<br>ITT | DB2114634<br>7.07 | Summary of On-treatment Drug-related Adverse Events | | SAC |

| Safety : | Safety : Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | 3.10 | Modified<br>ITT | DB2114634<br>7.07 | Summary of On-treatment Non-Serious Drug<br>Related Adverse Events | | SAC |
| 3.11. | 3.11 | Screen and<br>Run-in<br>Failure | DB2114634<br>7.09 | Summary of Pre-treatment Fatal Serious Adverse Events, Screen and Run-in Failure | | SAC |
| 3.12. | 3.12 | Screen and<br>Run-in<br>Failure | DB2114634<br>7.10 | Summary of Pre-treatment Non-Fatal Serious<br>Adverse Events, Screen and Run-in Failure | | SAC |
| 3.13. | 3.13 | Modified<br>ITT | DB2114634<br>7.11 | Summary of Pre-Treatment Non-Fatal Serious<br>Adverse Events, Modified Intent-to-treat | | SAC |
| 3.14. | 3.14 | Modified<br>ITT | DB2114634<br>7.12 | Summary of Fatal Serious Adverse Events | | SAC[1] |
| 3.15. | 3.15 | Modified<br>ITT | DB2114634<br>7.07 | Summary of Serious Adverse Events by System Organ Class | | SAC[1] |
| 3.16. | 3.16 | Modified<br>ITT | DB2114634<br>7.07 | Summary of Drug-Related Serious Adverse Events by System Organ Class | | SAC |
| 3.17. | 3.17 | Modified<br>ITT | DB2114634<br>7.13 | Summary of On-treatment Non-Fatal Serious<br>Adverse Events | | SAC |
| 3.18. | 3.18 | Modified<br>ITT | DB2114634<br>7.14 | Summary of Post-treatment Non- Fatal Serious Adverse Events | | SAC |
| 3.19. | 3.19 | Screen and<br>Run-in<br>Failure | DB2114634<br>7.15 | Summary of Pre-treatment Adverse Events<br>Leading to Withdrawal from the Study | | SAC |

| Safety : | Safety : Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.20. | 3.20 | Modified<br>ITT | DB2114634<br>7.16 | Summary of On-treatment Adverse Events Leading to Discontinuation of Study Treatment or Withdrawal from the Study | | SAC |
| 3.21. | 3.21 | Modified<br>ITT | DB2114634<br>7.17 | Summary of On-treatment Adverse Events of Special Interest | | SAC[1] |
| 3.22. | 3.22 | Modified<br>ITT | DB2114634<br>7.18 | Summary of Fatal Serious Adverse Events of Special Interest | | SAC |
| 3.23. | 3.23 | Modified<br>ITT | DB2114634<br>7.19 | Summary of On-treatment Non-Fatal Serious<br>Adverse Events of Special Interest | | SAC |
| 3.24. | 3.24 | Modified<br>ITT | DB2114634<br>7.20 | Summary of Fatal Drug Related Serious Adverse Events | | SAC |
| 3.25. | 3.25 | Modified<br>ITT | DB2114634<br>7.21 | Summary of On-treatment Non-Fatal Drug Related Serious Adverse Events | | SAC |
| 3.26. | 3.26 | Modified<br>ITT | DB2114634<br>7.22 | Summary of Chemistry Data | | SAC |
| 3.27. | 3.27 | Modified<br>ITT | DB2114634<br>7.23 | Summary of Change from Baseline in Chemistry Data | | SAC |
| 3.28. | 3.28 | Modified<br>ITT | DB2114634<br>7.24 | Summary of Chemistry Data Outside the Normal Range | | SAC |
| 3.29. | 3.29 | Modified<br>ITT | DB2114634<br>7.25 | Summary of Chemistry Changes from Baseline Relative to the Normal Range | | SAC |
| 3.30. | 3.30 | Modified<br>ITT | DB2114634<br>7.26 | Summary of Haematology Data | | SAC |

| Safety : | Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.31. | 3.31 | Modified<br>ITT | DB2114634<br>7.27 | Summary of Change from Baseline in Haematology Data | | SAC |
| 3.32. | 3.32 | Modified<br>ITT | DB2114634<br>7.28 | Summary of Haematology Data Outside the Normal Range | | SAC |
| 3.33. | 3.33 | Modified<br>ITT | DB2114634<br>7.29 | Summary of Haematology Changes from Baseline Relative to the Normal Range | | SAC |
| 3.34. | 3.34 | Modified<br>ITT | HZC113684<br>7.27 | Summary of Urinalysis Data | | SAC |
| 3.35. | 3.35 | Modified<br>ITT | DB2114634<br>7.30 | Summary of Vital Signs | | SAC |
| 3.36. | 3.36 | Modified<br>ITT | DB2114634<br>7.31 | Summary of Change from Baseline in Vital Signs | | SAC |
| 3.37. | 3.37 | Modified<br>ITT | DB2114634<br>7.32 | Statistical Analysis of Pulse Rate (bpm) | | SAC |
| 3.38. | 3.38 | Modified<br>ITT | DB2114634<br>7.33 | Statistical Analysis of Systolic Blood Pressure (mmHg) | | SAC |
| 3.39. | 3.39 | Modified<br>ITT | DB2114634<br>7.34 | Statistical Analysis of Diastolic Blood Pressure (mmHg) | | SAC |
| 3.40. | 3.40 | Modified<br>ITT | DB2114634<br>7.35 | Summary of ECG Values | | SAC |
| 3.41. | 3.41 | Modified<br>ITT | DB2114634<br>7.36 | Summary of Change from Baseline in ECG Values | | SAC |

| Safety : | Tables | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.42. | 3.42 | Modified<br>ITT | DB2114634<br>7.37 | Summary of QTc(F) (msec) Categories | | SAC |
| 3.43. | 3.43 | Modified<br>ITT | DB2114634<br>7.38 | Summary of Change From Baseline in QTc(F) (msec) Categories | | SAC |
| 3.44. | 3.44 | Modified<br>ITT | DB2114634<br>7.39 | Statistical Analysis of QTc(F) (msec) | | SAC |
| 3.45. | 3.45 | Modified<br>ITT | DB2114634<br>7.40 | Statistical Analysis of PR Interval (msec) | | SAC |
| 3.46. | 3.46 | Modified<br>ITT | DB2114634<br>7.41 | Statistical Analysis of ECG Heart Rate (bpm) | | SAC |
| 3.47. | 3.47 | Modified<br>ITT | DB2114634<br>7.42 | Summary of ECG Result Interpretations | | SAC |
| 3.48. | 3.48 | Modified<br>ITT | DB2114634<br>7.44 | Summary of All ECG Abnormalities | | SAC |

### 10.14.9. Safety Figures

| Safety | Safety : Figures | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 3.1. | 3.1 | Modified<br>ITT | DB2114634<br>7.01 | Scatter Plots of Maximum Post Baseline versus Baseline for<br>Chemistry Parameters with an Upper Limit of Normal Range | | SAC |
| 3.2. | 3.2 | Modified<br>ITT | DB2114634<br>7.02 | Box Plots of Change from Baseline to Maximum Post-baseline for Chemistry Parameters with an Upper Limit of Normal Range | | SAC |
| 3.3. | 3.3 | Modified<br>ITT | DB2114634<br>7.03 | Scatter Plots of Minimum Post Baseline versus Baseline for<br>Chemistry Parameters with a Lower Limit of Normal Range | | SAC |
| 3.4. | 3.4 | Modified<br>ITT | DB2114634<br>7.04 | Box Plots of Change from Baseline to Minimum Post-baseline for Chemistry Parameters with a Lower Limit of Normal Range | | SAC |
| 3.5. | 3.5 | Modified<br>ITT | DB2114634<br>7.05 | Scatter Plots of Maximum Post Baseline versus Baseline for Haematology Parameters with an Upper Limit of Normal Range | | SAC |
| 3.6. | 3.6 | Modified<br>ITT | DB2114634<br>7.06 | Box Plots of Change from Baseline to Maximum Post-baseline for Haematology Parameters with an Upper Limit of Normal Range | | SAC |
| 3.7. | 3.7 | Modified<br>ITT | DB2114634<br>7.07 | Scatter Plots of Minimum Post Baseline versus Baseline for Haematology Parameters with a Lower Limit of Normal Range | | SAC |
| 3.8. | 3.8 | Modified<br>ITT | DB2114634<br>7.08 | Box Plots of Change from Baseline to Minimum Post-baseline for Haematology Parameters with A Lower Limit of Normal Range | | SAC |
| 3.9. | 3.9 | Modified<br>ITT | DB2114634<br>7.09 | Trellis Display of Maximum Post-baseline versus Baseline for Liver Function Test Parameters | | SAC |
| 3.10. | 3.10 | Modified<br>ITT | DB2114634<br>7.10 | Least Squares Means Change from Baseline (95% CI) in Pre-dose Pulse Rate (bpm) | | SAC |

| Safety | Safety : Figures | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 3.11. | 3.11 | Modified<br>ITT | DB2114634<br>7.11 | Least Squares Means Change from Baseline (95% CI) in Pre-dose Systolic Blood Pressure (mmHg) | | SAC |
| 3.12. | 3.12 | Modified<br>ITT | DB2114634<br>7.12 | Least Squares Means Change from Baseline (95% CI) in Pre-dose Diastolic Blood Pressure (mmHg) | | SAC |
| 3.13. | 3.13 | Modified<br>ITT | DB2114634<br>7.13 | Empirical Distribution Function Plot of Maximum Post-baseline QTc(F) (msec) | | SAC |
| 3.14. | 3.14 | Modified<br>ITT | DB2114634<br>7.14 | Empirical Distribution Function Plot of Change from Baseline in Maximum Post-baseline QTc(F) (msec) | | SAC |
| 3.15. | 3.15 | Modified<br>ITT | DB2114634<br>7.15 | Least Squares Means Change from Baseline (95% CI) in Pre-dose QTc(F) (msec) | | SAC |
| 3.16. | 3.16 | Modified<br>ITT | DB2114634<br>7.16 | Least Squares Means Change from Baseline (95% CI) in Pre-dose PR Interval (msec) | | SAC |
| 3.17. | 3.17 | Modified<br>ITT | DB2114634<br>7.17 | Least Squares Means Change from Baseline (95% CI) in Pre-dose Heart Rate (bpm) | | SAC |

### 10.14.10. ICH Listings

| ICH: Listings | | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study P | opulation | | | | | |
| 1. | 1. | Screen and<br>Run in<br>Failure | ES7 | Listing of Reasons for Screen Failure / Run-in Failure | | SAC |
| 2. | 2. | Modified ITT | DB2114634<br>5.01 | Listing of Reasons for Withdrawal | | SAC |
| 3. | 3. | Modified ITT | DB2114634<br>5.02 | Listing of Planned and Actual Treatments | | SAC |
| 4. | 4. | Modified ITT | DV2 | Listing of Important Protocol Deviations | | SAC |
| 5. | 5. | Modified ITT | DV2 | Listing of Participants Excluded from PP population | | SAC |
| 6. | 6. | Modified ITT | DB2114634<br>5.03 | Listing of Inclusion, Exclusion or Randomisation Criteria Deviations | | SAC |
| 7. | 7. | Modified ITT | DB2114634<br>5.04 | Listing of Date of and Reason for Breaking Treatment Blind During the Study | | SAC |
| 8. | 8. | Modified ITT | DB2114634<br>5.05 | Listing of Demographic Characteristics | Birth date will be presented as 'YYYY' | SAC |
| 9. | 9. | Modified ITT | DB2114634<br>5.06 | Listing of Race | | SAC |
| 10. | 10. | Modified ITT | DB2114634<br>5.17 | Listing of COPD Concomitant Medications | | SAC |

| ICH : Lis | stings | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | Example Snell | | Programming Notes | Deliverable<br>[Priority] |
| 11. | | | DB2114634 Listing of Non-COPD Concomitant Medications 5.18 | | | SAC |
| 12. | 12. | Modified ITT | DB2114634<br>5.07 | Listing of Screening Lung Function Test Results | | SAC |
| Efficacy | 1 | • | | | | |
| 13. | 13. | Modified ITT | DB2114634<br>6.01 | Listing of Raw FEV1 (L) and FVC (L) | | SAC |
| Safety | | | | | • | |
| 14. | 14 Modified ITT DB2114634 | | DB2114634<br>7.01 | Listing of Exposure | | SAC |
| 15. | 15. | All Subjects<br>Enrolled | DB2114634<br>7.02 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 16. | 16. | All Subjects<br>Enrolled | DB2114634<br>7.03 | Listing of All Adverse Events | | SAC |
| 17. | 17. | All Subjects<br>Enrolled | AE2 | Listing of Relationship Between Adverse Event<br>System Organ Classes, Preferred Terms, and<br>Verbatim Text | | SAC |
| 18. | 18. | All Subjects<br>Enrolled | DB2114634<br>7.04 | Listing of Non-fatal Serious Adverse Events | | SAC |
| 19. | 19. | 19. All Subjects DB2114634 Listing of Fatal Adverse Events 7.05 | | | SAC | |
| 20. | 20. | All Subjects<br>Enrolled | DB2114634<br>7.06 | Listing of On-Treatment Drug Related SAEs | | SAC |

| ICH : Li | ICH : Listings | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 21. | 21. | Modified ITT | DB2114634<br>7.07 | Listing of Subject Numbers for On-treatment Adverse<br>Events of Special Interest | | SAC |
| 22. | 22. | All Subjects<br>Enrolled | DB2114634<br>7.08 | Listing of Adverse Events leading to Discontinuation of Study Treatment or Withdrawal from the Study | | SAC |
| 23. | 23. | Modified ITT | DB2114634<br>7.09 | Listing of Potential Investigational Product Inhaler Malfunctions Reported by Subjects | | SAC |
| 24. | 24. | Modified ITT | DB2114634<br>7.10 | Listing of Chemistry Values for Subjects with at Least One Value outside the Normal Range | | SAC |
| 25. | 25. | Modified ITT | DB2114634<br>7.11 | Listing of Haematology Values for Subjects with at Least One Value outside the Normal Range | | SAC |

## 10.14.11. Non-ICH Listings

| Non-ICI | Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study P | opulation | | | | | |
| 26. | 26. | All Subjects<br>Enrolled | DB2114634<br>5.08 | Listing of Reasons for Withdrawal- Subjects Randomised but Not in the Modified Intent-to-Treat Population | | SAC |
| 27. | 27. | All Subjects<br>Enrolled | DB2114634<br>5.10 | Listing of Treatment Misallocations | | SAC |
| 28. | 28. | Modified<br>ITT | DB2114634<br>5.11 | Listing of Medical Conditions | | SAC |
| 29. | 29. | Modified<br>ITT | DB2114634<br>5.12 | Listing of Past Cholecystectomies | | SAC |
| 30. | 30. | Modified<br>ITT | DB2114634<br>5.13 | Listing of Family History of Cardiovascular Risk Factors | | SAC |
| 31. | 31. | Modified<br>ITT | DB2114634<br>5.14 | Listing of COPD History | | SAC |
| 32. | 32. | Modified<br>ITT | DB2114634<br>5.15 | Listing of Smoking History and Smoking Status | | SAC |
| 33. | 33. | Modified<br>ITT | DB2114634<br>5.16 | Listing of mMRC Dyspnoea Scale | | SAC |
| 34. | 34. | Modified<br>ITT | DB2114634<br>5.19 | Relationship between ATC Level 1, Ingredient and Verbatim Text | | SAC |
| 35. | 35. | Modified<br>ITT | DB2114634<br>5.20 | Listing of Treatment Compliance Data | | SAC |

| Non-ICI | H : Listings | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 36. | 36. | All Subjects<br>Enrolled | DB2114634<br>5.21 | Listing of All Protocol Deviations | | SAC |
| Efficacy | У | | | | | |
| 37. | 37. | Modified<br>ITT | DB2114634<br>6.02 | Listing of Derived FEV1 Endpoints | | SAC |
| 38. | 38. | Modified<br>ITT | DB2114634<br>6.03 | Listing of Derived FVC Endpoints | | SAC |
| 39. | 39. | Modified<br>ITT | DB2114634<br>6.04 | Listing of BDI/TDI | | SAC |
| 40. | 40. | Modified<br>ITT | DB2114634<br>6.05 | Listing of SGRQ Scores | | SAC |
| 41. | 41. | Modified<br>ITT | DB2114634<br>6.06 | Listing of Derived Rescue Endpoints | | SAC |
| 42. | 42. | Modified<br>ITT | DB2114634<br>6.07 | Listing of CAT Scores | | SAC |
| 43. | 43. | Modified<br>ITT | DB2114634<br>6.08 | Listing of COPD Exacerbations | | SAC |
| 44. | 44. | Modified<br>ITT | Non-Standard<br>EFF_L1 | Listing of Healthcare Resource Utilisation | | SAC |
| Safety | | | | | | |
| 45. | 45. | Modified<br>ITT | DB2114634<br>7.12 | Listing of Immunology Data for subjects with at least one Reactive Result | | SAC |

| Non-ICH: Listings | | | | | | |
|---|---|---|---|---|---|---|
| IMCT<br>No. | China<br>Subgroup<br>No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 46. | 46. | Modified<br>ITT | DB2114634<br>7.13 | Listing of Virology Data | | SAC |
| 47. | 47. | Modified<br>ITT | DB2114634<br>7.14 | Listing of Urinalysis Data | | SAC |
| 48. | 48. | Modified<br>ITT | DB2114634<br>7.15 | Listing of Vital Signs | | SAC |
| 49. | 49. | Modified<br>ITT | DB2114634<br>7.18 | Listing of ECG Values for Subjects with Any Abnormal ECG Interpretation | | SAC |
| 50. | 50. | Modified<br>ITT | DB2114634<br>7.19 | Listing of ECG Findings for Subjects with Any Abnormal ECG Interpretation | | SAC |
| 51. | 51. | Modified<br>ITT | DB2114634<br>7.20 | Listing of Liver Event Results and Time of Event Relative to Treatment | | SAC |
| 52. | 52. | Modified<br>ITT | DB2114634<br>7.21 | Listing of Liver Event Information for RUCAM Score | | SAC |
| 53. | 53. | Modified<br>ITT | DB2114634<br>7.22 | Listing of Liver Biopsy Details | | SAC |
| 54. | 54. | Modified<br>ITT | DB2114634<br>7.23 | Listing of Liver Imaging Details | | SAC |

#### 10.15. Appendix 15: Example Mock Shells for Data Displays

Example : EFF\_L1 Page 1 of n

Protocol : AC4117410 Population : ITT

Listing 41
Listing of Healthcare Resource Utilisation

| Investigator at<br>Centre/<br>Subject | Date<br>of Contact | Number of office/practice visits | Number of urgent<br>care/outpatient<br>Visits | Number of emergency room visits | Number of days in intensive care | Number of days<br>in general ward | Was this contact<br>due to an<br>exacerbation |
|---|---|---|---|---|---|---|---|
| PPD | 21May2013<br>01MAY2013 | 0 | 1 | 0 | 0 | 0 | N |